

Study Number: KIN-1901-2001

Study Title: A Multi-Center, Adaptive, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of Gimsilumab in Subjects With Lung Injury or Acute Respiratory Distress Syndrome (ARDS) Secondary to Coronavirus Disease 2019 (COVID-19)

Statistical Analysis Plan

Version 4, 17-November-2020

NCT04351243

# **PAREXEL International**

Kinevant

KIN-1901-2001

A Multi-Center, Adaptive, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of Gimsilumab in Subjects With Lung Injury or Acute Respiratory Distress Syndrome (ARDS) Secondary to Coronavirus Disease 2019 (COVID-19)

# **Statistical Analysis Plan**

Version: 4.0

**PAREXEL Project Number: 250621** 

# **SPONSOR SIGNATURE PAGE**

| Approved by: | | |
|--------------|------------------------------------|-------------|
| | On Behalf of Kinevant Sciences Inc | <b>Date</b> |
| | On Behalf of Kinevant Sciences Inc | Date |
| | Kinevant Sciences Inc | Date |

# PAREXEL SIGNATURE PAGE

Signature(s) below confom that the Statistical Analysis Plan was developed in accordance with SOP-GDO-WW-019 and that it is approved for release.

This document has been approved and signed electronically on the final page by the following:

| | Signatory |
|--------|-----------|
| Author | |

# TABLE OF CONTENTS

| 1 | INTRODUCTION | . 10 |
|---|---|---|
| 2 | STUDY OBJECTIVES | . 11 |
| 2.1 | Primary Objective(s) | . 11 |
| 2.2 | Secondary Objective(s) | . 11 |
| 2.3 | Exploratory Objective(s) | . 11 |
| 3 | INVESTIGATIONAL PLAN | . 12 |
| 3.1 | Overall Study Design and Plan | . 12 |
| 3.2 | Database locks | . 13 |
| 3.3 | Determination of Sample Size | . 13 |
| 3.4 | Endpoints | . 14 |
| 3.4.1 | 1 Efficacy Variables | . 14 |
| 3.4.2 | 2 Safety Variables | . 14 |
| 3.5 | Exploratory Variables | . 15 |
| 4 | STATISTICAL METHODS | . 16 |
| 4.1 | Data Quality Assurance | . 16 |
| 4.2 | General Presentation Considerations | . 16 |
| 4.2.1 | 1 Study Periods | . 16 |
| 4.2.2 | 2 Study Visits and Windowing | . 17 |
| 4.2.3 | 3 Missing dates | . 18 |
| 4.2.4 | 4 Conventions | . 18 |
| 4.3 | Software | . 19 |
| 4.4 | Study Subjects | . 19 |
| <b>4.4.</b> 1 | 1 Disposition of Subjects | . 19 |
| 4.4.2 | 2 Protocol Deviations | . 19 |
| 4.5 | Analysis Sets | . 19 |
| 4.6 | Demographic and Other Baseline Characteristics | . 20 |
| 4.7 | Prior, Concomitant, and Prohibited Medications and Procedures | . 21 |
| 4.8 | Efficacy Evaluation | . 22 |
| 4.8.1 | 1 Analysis and Data Conventions | . 22 |
| 4.8.1 | | |
| 4.8.1 | 1.2 Adjustments for Covariates | . 22 |
| 4.8.1 | 1.3 Handling of Dropouts or Missing Data | . 22 |
| 4.8.1 | 1.4 Multiple Comparisons/Multiplicity | . 22 |
| 4.8.1 | 1.5 Examination of Subgroups | . 23 |
| 4.8.1 | | . 24 |
| 4.8.1 | | |
| 4.8. | | |
| 4.8.1 | | |
| 4.8. | | |
| 4.8.1 | · | |
| 4.8. | | |
| 4.8. | | |
| 4.8. | | |
| 4.8.2 | | |

**Project Document Effective Date**: Date of last signature 

# PAREXEL International

| Kinevant<br>KIN-1901-2001 | Statistical Analysis Plan |
|---|---|
| 4.8.3 Key Secondary Efficacy Analysis | |
| 4.8.3.1 Survival and no mechanical ventilation on Day 29 | |
| 4.8.3.2 Mechanical ventilation-free days by Day 29 | |
| 4.8.3.3 Time to hospital discharge | |
| 4.8.4 Other Secondaiy and Exploratory Efficacy Analyses | 35 |
| 4.9 Safety Evaluation | 39 |
| 4.9.1 Extent of Exposure | 39 |
| 4.9.2 Adverse Events | 39 |
| 4.9.2.1 AE Summaries by system organ class (SOC) and prefened tenn | (PT)40 |
| 4.9.2.2 AE of Special Interest (AESI) | 41 |
| 4.9.2.3 Adverse event listings | 41 |
| 4.9.3 Clinical Laboratory Evaluation | 41 |
| 4.9.4 Vital Signs, Physical Findings and Other Observations Related to | Safety43 |
| 4.9.5 Independent Data Monitoring Committee | 44 |
| 4.10 Other Analyses | |
| 4.10.1 Pha11nacokinetics | 45 |
| 4.10.2 hnmunogenicity | 45 |
| 4.10.3 Biomarker | 45 |
| 4.11 Changes <b>in</b> the Conduct of the Study or Planned Analysis | 46 |
| 5 INTERIM ANALYSES | 47 |
| 5.1 Interim Analysis 1 | 47 |
| 5.1.1 Subjects to be included in interim analysis 1 | 47 |
| 5.1.2 Analysis of efficacy endpoints at interim analysis 1 | 47 |
| 5.1.3 Futility criteria at interim analysis 1 | 47 |
| 5.2 Interim Analysis 2 | |
| 5.2.1 Subjects to be included in interim analysis 2 | |
| 5.2.2 Analysis of efficacy endpoints at interim analysis 2 | |
| 5.2.3 Superiority stopping criteria at interim analysis 2 | |
| 5.2.4 Futility stopping criteria at interim analysis 2 | |
| 5.2.5 Sample size re-estimation at interim analysis 2 | 48 |
| 5.2.6 Interim analysis 2 outcome | |
| 6 REFERENCES | 50 |
| 7 APPENDICES | 51 |
| 7.1 Schedule of Assessments | 52 |
| 7.2 Adverse Events of Special Interest. | 56 |

Related to: SOP-GDO-WW-019 

# **REVISION HISTORY**

| Version No. | Effective Date | Summary of Change(s) |
|---|---|---|
| 0.1 | 06Apr2020 | New document |
| 0.2 | 15Apr2020 | Incorporate Parexel internal review comments |
| 0.3 | 19Apr2020 | Incorporate Sponsor statistical review comments |
| 0.4 | 24Apr2020 | Incorporate Sponsor review comments |
| 0.5 | 01May2020 | Incorporate Sponsor review comments |
| 1.0 | 06May2020 | Final version for signature |
| 1.1 | 19Jun2020 | Update to align with Protocol v4.0 (12Jun2020) and to |
| | | address FDA comments on SAP v1.0. Major updates: |
| | | - Updates to key secondary endpoints. |
| | | - Change missing data imputation method from LOCF |
| | | to tipping point method. |
| | | - Use estimand framework to describe primary and key secondary efficacy analyses. |
| 1.2 | 21Jun2020 | Incorporate Sponsor statistical review comments |
| 1.3 | 22Jun2020 | Additional details for interim analysis and missing data |
| | | analyses added. |
| 2.0 | 26Jun2020 | Incorporate final Sponsor review comments. Final version for |
| | | signature |
| 2.1 | 20Jul2020 | Incorporate FDA comments on SAP v2. and editorial changes |
| | | to fix minor typographical errors and add clarity. |
| 2.2 | 11Aug2020 | Add superiority boundary for IA2, incorporate Parexel |
| 2.0 | 124 2020 | internal review comments |
| 3.0 | 12Aug2020 | Incorporate final comments. Final version for signature. |
| 3.1 | 19Oct2020 | Update per IA2 decisions: - Section 4.7 – Add summaries of any steroid use, any dexamethasone use, any other COVID-19 therapies. |
| | | - Section 4.8.1.5 – Add new subgroup 'Baseline |
| | | invasive ventilator use or severe ARDS at baseline' |
| | | - Section 4.8.4 – Amend proposed analyses for 7-point |
| | | ordinal scale to include shift tables and remove odds |
| | | ratios and CMH tests. |
| | | - Add section 5.2.6: Interim analysis 2 outcome |
| 3.2 | 30Oct2020 | Incorporate sponsor comments. Add multi-state competing |
| | | risks analysis as supplementary analysis for time to hospital |
| | | discharge and time to clinical improvement (section 4.8.1.13). |
| 4.0 | 13Nov2020 | Incorporate final comments. Final version for signature. |

TP-GDO-WW-016-07.a CO
Effective Date: 30 Jan 19
Related to: SOP-GDO-WW-019

# LIST OF ABBREVIATIONS

| Abbreviation / Acronym | Definition / Expansion |
|------------------------|-----------------------------------------------|
| ADA | Anti-drng antibodies |
| AE | Adverse event |
| AESI | Adverse events of special interest |
| ALP | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| ANCOVA | Analysis of covariance |
| aPTT | Activated partial thromboplastin time |
| ARDS | Acute respiratory distress syndrome |
| AST | Aspartate aminotransferase |
| BILI | Total bilirnbin |
| BMI | Body Mass Index |
| BP | Blood pressure |
| CI | Confidence interval |
| CMH | Cochran-Mantel-Haenszel |
| CMQ | Company MedDRA que1y |
| COVID-19 | Coronavims disease 2019 |
| CPAP | Continuous positive aiiway pressure |
| CRP | C-reactive protein; |
| DBP | Diastolic blood pressure |
| DMC | Data monitoring committee |
| DoD | Day-of-discharge |
| DRM | Data Review Meeting |
| EAIR | Exposure-adjusted incidence rate |
| ECMO | Extracolporeal membrane oxygenation |
| eCRF | Electronic Case Repoli Folm |
| eGFR | Estimated glomernlar filtration rate |
| EoS | End-of-study |
| ET | Early telmination |
| FAS | Full analysis set |
| FiO2 | Fraction of inspii ed oxygen |
| TP-GDO-WW-016-07 a | CONFIDENTIAL Project Document Version No. 4.0 |

TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

**Project Document Effective Date:** Date ofla.st signature


| Abbreviation / Acronym | Definition / Expansion |
|------------------------|--------------------------------------------------|
| GM-CSF | Granulocyte macrophage-colony stimulating factor |
| HR | Heart rate |
| IA | Interim analysis |
| ICU | Intensive care unit |
| ITT | Intent-to-ti·eat |
| IV | Inti-avenous |
| LDH | Lactate dehydrogenase |
| LIS | Lung injmy score |
| LOCF | Last observation calTied fo1ward |
| LVEF | Left venti-icular ejection fraction |
| MDRD | Modification of Diet in Renal Disease |
| MMRP | Mixed model with repeated measures |
| MedDRA | Medical Dictionaly for Regulatoly Activities |
| NA | Not available |
| NEWS | National Early Warning Score |
| 02 | Oxygen |
| PEEP | Positive end-expiratory pressure |
| PIF | PaOi/Fi02 ratio |
| Pa02 | Paiiial pressure of oxygen |
| PCR | Polymerase chain reaction |
| P-D | Patient days |
| PK | Phannacokinetics |
| pp | Per-protocol |
| PT | Prefe1Ted Tenn |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SARS-CoV-2 | Severe acute respiratory syndrome corona vims 2 |
| SBP | Systolic blood pressure |
| SD | Standard deviation |
| SMQ | Standard MedDRA que1y |
| soc | System Organ Class |

TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

Project Document Effective Date: Date ofla.st signature


# PAREXEL International

| Kinevant |
|---------------|
| KIN-1901-2001 |

Statistical Analysis Plan

| Abbreviation / Acronym | Definition / Expansion |
|------------------------|----------------------------------------------------|
| SOFA | Sequential Organ Failure Assessment |
| SP-D | Surfactant protein D |
| SpO2 | Peripheral capillary oxygen saturation |
| TEAE | Treatment-emergent adverse event |
| TLF | Tables, Listings, Figures |
| WHODDE | Wodd Health Organization - Dmg Dictionary Enhanced |

## 1 INTRODUCTION

In December 2019, the city of Wuhan, China experienced an outbreak of coronavirus disease 2019 (COVID-19), caused by a novel coronavirus, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). As of March 2020, COVID-19 has become a global pandemic, and there are currently no approved agents available to treat coronaviruses. SARS-CoV-2 infection often induces an overactive immune response that causes significant lung damage, leading to acute respiratory distress syndrome (ARDS) and ultimately death. Granulocyte macrophage-colony stimulating factor (GM-CSF), a hematopoietic growth factor and immunomodulatory cytokine, is believed to have a key driver of cytokine storm and lung hyper-inflammation. Targeting GM-CSF using an anti-GM-CSF antibody, gimsilumab (KIN-1901), represents a promising strategy to treat patients who have developed lung injury or ARDS secondary to COVID-19.

KIN-1901-2001 is a randomized, double-blind, placebo-controlled study of gimsilumab for the treatment of lung injury or ARDS secondary to COVID-19. A total of 270 subjects are planned to be treated with IV gimsilumab on day 1 (400mg) and day 8 (200mg) or matching IV placebo (saline solution on days 1 and 8). This study consists of a 2-week Treatment Period and a 22-week Follow-up Period.

This study will have two database locks, the first when all subjects have completed through Day 43 or withdraw from the study early or meet the primary mortality endpoint. The second database lock will be when the last subject completes the Day 169/End-of-study (EoS) visit.

This statistical analysis plan (SAP) provides a detailed description of the statistical methods and analyses to be carried out in support for study KIN-1901-2001.

The following will be collected and not entered into the clinical study database until the database is locked:

- Pharmacokinetic data
- Immunogenicity data
- Exploratory biomarkers

The analyses described in this SAP are based upon the following study documents:

- Study Protocol, Version 2.0 (April 5, 2020)
- Study Protocol, Version 5.0 (August 17, 2020)
- KIN-1901-2001 DMC Charter Version 3.1 (July 11, 2020)
- eCRF (September 29, 2020)

#### 2 STUDY OBJECTIVES

# 2.1 Primary Objective(s)

The primary objective is to evaluate the impact of intravenous (IV) treatment with gimsilumab on mortality in subjects with lung injury or ARDS secondary to COVID-19.

# 2.2 Secondary Objective(s)

Key Secondary Objectives:

- To assess the effect of gimsilumab on ventilation requirements
- To assess the effect of gimsilumab on overall duration of hospitalization

## Additional Secondary Objectives:

- To assess the effect of gimsilumab on the need for Intensive Care Unit (ICU) level of care
- To assess the effect of gimsilumab as measured by the National Early Warning Score (NEWS)
- To assess the effect of gimsilumab as assessed by the Sequential Organ Failure Assessment (SOFA) score
- To assess the effect of gimsilumab as measured by the 7-point ordinal scale
- To assess the effect of gimsilumab on peripheral capillary oxygen saturation / fraction of inspired oxygen (SpO<sub>2</sub>/FiO<sub>2</sub>)
- To assess the effect of gimsilumab on oxygenation requirements
- To assess changes in on-treatment viral load
- To assess the effect of gimsilumab on biomarkers of inflammation
- To determine the pharmacokinetic (PK) properties of gimsilumab
- To assess the immunogenicity of gimsilumab
- To determine the safety and tolerability of gimsilumab

# 2.3 Exploratory Objective(s)

- To explore the effect of gimsilumab on serum cytokine concentrations and surfactant protein D (SP-D)
- To explore the effect of gimsilumab on other measurements of lung injury that may be performed during standard care (e.g., Lung Injury Score [LIS], chest radiography, PaO<sub>2</sub>/FiO<sub>2</sub> [P/F ratio], need for extracorporeal membrane oxygenation [ECMO])
- To explore the effect of gimsilumab on cardiac function (if measured)
- To assess the effect of gimsilumab on renal function

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant KIN-1901-2001

Statistical Analysis Plan

#### 3 INVESTIGATIONAL PLAN

# 3.1 Overall Study Design and Plan

This is a randomized, adaptive, double-blind, placebo-controlled study in male and/or female subjects who are at risk of developing, or have developed, ARDS consequent to moderate to severe COVID-19. This study will include subjects with moderate-to-severe disease. There will be 2 treatment aims, one receiving blinded gimsilumab, and one receiving blinded placebo.

Efficacy, safety, tolerability, phannacokinetics, and phaimacodynamics of gimsilumab will be assessed in hospitalized adult subjects diagnosed with COVID-19. Randomization will bestratified by:

- Subject's clinical status at Baseline
  - o Lung injmy/mild ARDS
  - o Moderate/severe ARDS

Lung injmy is defined as (1) requiring supplemental oxygen >4L 02 to maintain >92% SpO2, or (2) PaOi/FiO2:S 300 rmnHg (can be imputed).

ARDS is defined (ARDS Definition Task Force 2012) as:

- Bilateral opacities not fully explained by effusions, lobai lung collapse, or nodules;
- Respiratoly failme not fully explained by cai diac failw-e or fluid overload;
- Need objective assessment (e.g., echocai·diography) to exclude hydrostatic edema if no risk factor present.
- ARDS severity categories are defined as:
  - o Mild: 200 m1nHg, < PaOi/FiO2, :S300 rmnHg with PEEP or CPAP::::5 cm H2O.
  - o Moderate: 100 mmHg, < PaOi/FiO2, :S 200 rmnHg with PEEP::::5 cm H2O.
  - o Severe: PaOi/FiO2:Sl00 rmnHg with PEEP::::5 cm H2O.

A schematic of the study design is presented in <u>Figure 3-1</u>. Subjects will be assessed daily while hospitalized. Follow-up assessments are planned through Week 24, for a total study duration post-randomization of approximately 169 days (24 weeks). Follow-up visits at Days 15, 22, 29, 36, 43, 85 and 169 will be perfonned by phone if the subject has been discharged from the hospital. All subjects will undergo a series of efficacy, safety, and laboratoly assessments as detailed in the Schedule of Assessments (<u>Appendix 7.1</u>).

Each subject will palticipate for approximately 24 weeks, with a 2-week Treatment Period (last dose on Day 8) and a 22-week Follow-up Period. Treatment Anns for KIN-1901-2001:

**Arm 1:** Gimsilumab (400 mg) as a single IV infusion on Day 1 followed by a single 200 mg IV infusion on Day 8\* (N=135)

**Arm 2:** Placebo (0.9% saline solution) IV infusion on Day 1 and Day 8\* (N=135)

\*The Day 8 dose will be omitted if the subject is discharged from the hospital or is no longer in need of supplemental oxygen or ventilatory suppolt for >48 hours.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant

KIN-1901-2001 Statistical Analysis Plan

Asufficient number of subjects will be emolled to achieve approximately 270 evaluable subjects total, with 135 subjects per treatment aim. There will be two intelim analyses (IA):

1st IA: For safety and futility when 60 subjects have completed treatment and completed through study Day 15

**2<sup>nd</sup>** IA: For safety, superiority, and futility when 100 subjects have completed the study Day 29 Visit (for non-moltality endpoints) or have died (moltality data) by Day 43 (see Section 5.2.1 for details). The sample size re-estimation will be perfolmed to maintain the conditional power of 80% the primary analysis of M01 tality by Day 43.

Figure 3-1: Study Schematic



ARDS = acute respirato1y distress syndrnme; CRP = C-reactive prntein; EoS = End of Study; IV = intravenous; ICU = Intensive Care Unit; NEWS= National Early Warning Score; SOFA= Sequential Organ Failure Assessment

#### 3.2 Database locks

The database will be locked first when all subjects complete the Day 43 Visit, discontinue from the study eai·ly, or meet the primary m01tality endpoint. The second lock will occm when the last subject completes the Day 169/ EoS visit, discontinue from the study eai·ly, or died up to Day 169. Study unblinding will occm at the first database lock.

All analyses described in this SAP will be perfo1med at the 1<sup>st</sup> database lock. For the 2<sup>nd</sup> lock, all safety analyses will be perfo1med but efficacy analyses without new data (*e.g.* assessments only collected dming hospitalization if all subjects have been discharged by 1<sup>st</sup> database lock) may not be perfo1med again.

#### 3.3 Determination of Sample Size

There will be 270 subjects (135 subjects per treatment aim) with 1:1 randomization.

The comparisons between the treatment anns will have approximately 83% power and overall two-sided alpha level 0.05 (the equivalent one-sided overall significance level 0.025 will be used in the remainder of this SAP) to demonstrate a statistically significant reduction in moltality by Day 43 for

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

## PAREXEL International

Kinevant

KIN-1901-2001 Statistical Analysis Plan

gimsilumab compared to placebo when assuming tme propoltions of 15% and 30%, respectively and a superiolity / futility intelim analysis as described in <u>Section 5.2</u>.

The study will emoll at least 40%, but no more than 60%, of total patients in each of the 2 categories of clinical status: ([lung injmy/mild ARDS] or [moderate/severe ARDS]) at Baseline, which will be used as the stratified factor in the randomization.

# 3.4 Endpoints

# 3.4.1 Efficacy Variables

#### Primary:

• Mo1tality by Day 43

# Key Secondary:

- Propoltion of subjects who survived and not requiring mechanical ventilation on Day 29
- Mechanical ventilation-free days by Day 29
- Time to hospital discharge

#### Additional Secondary:

- Mortality by Days 15, 22, 29, 85, and 169 (EoS)
- Proportion of subjects who survived and were not requiring mechanical ventilation on Days 15, 22, and 43
- Mechanical ventilation-free days for all subjects by Days 15, 22, and 43.
- ICU-free days for all subjects by Days 15, 22, 29, and 43
- Incidence of mechanical ventilation use for all subjects Days 15, 22, 29, and 43.
- Incidence of ICU use for all subjects Days 15, 22, 29, 43
- Time to death by Day 43 and Day 169 (EoS)
- NEWS assessed daily while hospitalized
- SOFA score and each of the components assessed daily while in the ICU
- Status on the 7-point ordinal scale daily while hospitalized and on Days 15, 22, 29, 36, 43, 85, and 169 if discharged
- Time to clinical improvement
- Change from Baseline in SpOi/Fi02 assessed daily while hospitalized
- Incidence and duration of oxygen use during the study
- Change from Baseline in viral load as measured by quantitative polymerase chain reaction (PCR) test on Days 2, 9, and Day-of-discharge (DoD)
- Change from Baseline in D-dimer, cardiac troponin I, lactate dehydrogenase (LDH), fenitin, procalcitonin, and C-reactive protein (CRP) on Days 4, 8, and DoD (and Days 15, 22, 29, 36, and 43 if hospitalized)
- Selum gimsilumab concentrations on Days 1, 8, and DoD
- Anti-gimsilumab antibodies (ADAs) on Day 1 and DoD (and Days 15, 29, and 43 if hospitalized)

#### 3.4.2 Safety Variables

- Physical examinations
- Vital signs (supine blood pressure [BP] and pulse, oral body temperature, respiratoly rate)

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant KIN-1901-2001 Statistical Analysis Plan

- Clinical laboratory tests (hematology, clinical chemistry, and urinalysis parameters)
- Adverse event (AE) assessments
- Concomitant medication assessments

The above safety variables will be summarized by Day 43 and Day 169/EoS.

#### 3.5 **Exploratory Variables**

- Change from Baseline in the cytokine panel on Days 4, 8, and DoD (and Days 15 and 29 if hospitalized)
- Change from Baseline in LIS (if performed) daily while hospitalized
- Change from Baseline in chest radiographic assessment (if performed)
- Change from Baseline in P/F ratio (if performed) daily while hospitalized
- Incidence and duration of ECMO use
- Change from Baseline in left ventricular ejection fraction (LVEF) (when measured)
- Change from Baseline in eGFR [Modification of Diet in Renal Disease (MDRD) equation], assessed when central clinical safety laboratory measurements are collected during hospitalization

TP-GDO-WW-016-07.a **CONFIDENTIAL Project Document Version No. 4.0** Effective Date: 30 Jan 19 **Project Document Effective Date**: Date of last signature Related to: SOP-GDO-WW-019

#### 4 STATISTICAL METHODS

# 4.1 Data Quality Assurance

All tables, figures and data listings to be included in the report will be independently checked for consistency, integrity and in accordance with standard Parexel procedures.

#### 4.2 General Presentation Considerations

### 4.2.1 Study Periods

This study has two periods, the treatment period and the follow-up period (Figure 3-1). The follow-up period will be divided into two for analysis purposes, the first for follow-up through Day 43 and the second for Day 44 through the end-of study. Some assessments will only be done while subjects are hospitalized as detailed in the schedule of assessment (Appendix 7.1), because of this some endpoints during each period will not be available for all subjects. The hospitalization period will contain all assessments during either the treatment period or follow-up period that occur before the subject is discharged. The discharge period will cover the time starting the day after hospital discharge through the end-of-study. Differences in time at risk will also be taken to account at the endpoint level and each endpoint be analyzed using methods appropriate to its planned collection pattern. Medical events and medications will be classified into study periods using their start dates.

The following definitions will be applied:

**Treatment period (Day 1 – Day 15):** Starts on *first dose date* and ends at the earliest of *first dose date* + 14 and *end of study date*.

**Follow-up period 1 (Day 16 through Day 43):** Starts on *first dose date* + 15 and ends at the *Day 43 Visit date*.

**Follow-up period 2 (Day 44+):** Starts on *first dose date* + 43 and ends at the *end of study date*.

**Overall:** Treatment period, follow-up period 1 and follow-up period 2 combined.

**Overall - Hospitalized:** Study Day 1 to *date of discharge*. This period will include all assessments that were taken while the subject was hospitalized.

Overall – After Discharge: Day of discharge through end of study. This period starts at date of discharge + 1 and ends at the end of study date.

#### Where,

First dose date: Day 1, date first dose of study drug received.

End of study date: date of End-of-Study visit (Day 169/ EoS) if subject completes the study or date of early withdrawal if subject discontinues early or date of death.

**Date of discharge:** date subject is discharged from the hospital.

**Study Day:** <Assessment Date> - *first dose date* + 1 if <Assessment Date> is on or after *first dose date*. <Assessment Date> - *first dose date*, if <Assessment Date> is before *first dose date*.

Study drug: gimsilumab or placebo

**Study treatment:** administration of study drug on Day 1 and Day 8 (as required per protocol).

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant KIN-1901-2001

Statistical Analysis Plan

#### 4.2.2 Study Visits and Windowing

**Baseline:** the last available pre-ti-eatment assessment. All assessments should have time collected. If time is not collected and date of assessment is the same as the *first dose date*, then assessment will be assumed to be collected prior to ti-eatment unless schedule of assessments and protocol indicate planned collection is always after dosing.

**Day-of-Discharge (DoD):** day when subject is discharged from the hospital.

Early Termination (ET): day when subject withdraws from the study before completion.

**End-of-Study (EoS):** the end of study visit is at Day 169 (24 weeks after first dose) for subjects who complete the study.

#### **Study Visits:**

Planned study visits are detailed in <u>Table 4-1</u> and in the Schedule of Assessments (<u>Appendix 7.1</u>). Planned study visits that occur outside of their protocol defined window will be analyzed as repolied and there will no attempt to colTect visits that fall outside their planned time frame by applying analysis visit windows. Unscheduled visits will be assigned to a study visit if they fall into the study windows. Unscheduled visits that do not fall into scheduled study visit window will be included when classifying endpoints across a period (e.g. maximum value during study period) but will not be repolied in by visit summaries.

fu the case of multiple assessments on the same visit the following rnles will apply:

- If more than one assessment occurs during the same nominal visit time window of the planned visit, select the record closest to the nominal day for that paiiicular visit day.
- If there ai e two assessments that are equidistant from the nominal planned visit day, the data of the assessment after the scheduled study day will be used.
- If multiple measurements are all taken on the same day the earliest measurement of this day will be used.

**Table 4-1: Study Visit Windowing** 

| Visit | Study Day/Week | Window |
|-----------|----------------|------------|
| Screening | -7 to 1/0 | None |
| Baseline | 1/0 | None |
| Day2 | 2/1 | +/- 1 day* |
| Dav3 | 3/1 | +/- 1 day* |
| Dav4 | 4/1 | +/- 1 day* |
| Day5 | 5/1 | +/- 1 day* |
| Day6 | 6/1 | +/- 1 day* |
| Dav7 | 7/1 | +/- 1 day* |
| Dav8 | 8/2 | +/- 1 dav* |
| Day9 | 9/2 | +/- 1 day* |
| Dav 10 | 10/2 | +/- 1 day* |
| Dav 11 | 11/2 | +/- 1 dav* |
| Day 12 | 12/2 | +/- 1 day* |
| Dav 13 | 13/2 | +/- 1 day* |
| Dav 14 | 14/2 | +/- 1 day* |
| Day 15 | 15/2 | +/- 2 day |

TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL

**Project Document Version No. 4.0** 

**Project Document Effective Date:** Date of last signature


Kinevant

KIN-1901-2001 Statistical Analysis Plan

| Visit | Study Dav/Week | Window |
|-------------|----------------|-----------|
| Dav22 | 22/3 | +/- 2 dav |
| Day29 | 29/4 | +/- 2 day |
| Dav36 | 36/5 | +/- 2 day |
| Dav43 | 43/6 | +/- 2 day |
| Day85 | 85/12 | +/- 2 day |
| Dav 169/EoS | 169/24 | +/- 2 day |

<sup>\*</sup>no window will be applied for assessments collected daily during hospitalization per Schedule of Assessments (Aooendix 7.1)

# 4.2.3 Missing dates

Every effolt will be made to collect complete dates for all study assessments. The following date imputation rules will be applied for missing or paltial dates:

- If month and year available, set start date to latest of (1<sup>st</sup> of the *month,first dose date*), if end date is complete and imputed strut date > end date, set imputed strut date to end date 1.
- If year available: Set strut date to Janualy 1<sup>st</sup> of year recorded, if end date is complete and imputed strut date > end date, set imputed strut date to end date 1.
- If strut date is completely missing, set to *first dose date*, if end date is complete and imputed strut date > end date, set imputed strut date to end date- 1.
- If any imputed date results in an improbable date (e.g. date occurs in the future, date occurs after subject died), set to *first dose date*.

#### 4.2.4 Conventions

Continuous data will be summarized in tenns of the mean, standai deviation (SD), median, minimum, maximum, and number of observations, unless othelwise stated. Continuous data that are expected to be skewed will be presented in tenns of the maximum, upper quaitile, median, lower qurutile, minimum, and number of observations. The minimum and maximum will be repolted to the same number of decimal places as the raw data recorded in the database. The mean, median, lower qurutile, and upper quaitile will be repolted to one more decimal place than the raw data recorded in the database. The SD will be repolted to two more decimal places than the raw data recorded in the database. In general, the maximum number of decimal places repolted shall be four for any summary statistic.

Categorical data will be smnmru ized in tenns of the number of subjects providing data at the relevant time point (n), frequency counts and percentages. Any planned collapsing of categories will be detailed in the SAP text and the data displays.

Percenta ges will be presented to one decimal place. Percenta ges will not be presented for zero counts. Percenta ges will be calculated using n as the denominator. If sample sizes ai e small, the data displays will show the percentages, but any textual report will describe frequencies only.

Changes from baseline in categorical data will be summarized using shift tables where appropriate.

P-values greater than or equal to 0.001, in general, will be presented to three decimal places. P-values less than 0.001 will be presented as "<0.001".

Confidence intervals will be presented to one more decimal place than the raw data.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant KIN-1901-2001

Statistical Analysis Plan

#### 4.3 Software

All report outputs will be produced using SAS® version 9.4 or a later version in a secure and validated environment.

# 4.4 Study Subjects

# 4.4.1 Disposition of Subjects

A clear accounting of the disposition of all subjects who enter the study will be provided, from screening to study completion.

#### Summaries will include:

- the number of subjects randomized (full analysis set)
- the number and percentage of subjects treated (with any amount of study drug)
- the number and percentage of subjects entering, withdrawing from study treatment, withdrawing from the study and completing each phase of the study by treatment group and overall. Withdrawals from the study and from study treatment will also be summarized by major reason. (Analysis set: Full Analysis Set)

By-subject listings of eligibility details, randomization details, visit dates and withdrawal/study completion details (including reason for discontinuation and duration of treatment prior to discontinuation) will be provided.

#### 4.4.2 Protocol Deviations

Major protocol deviations are defined as those deviations from the protocol likely to have an impact on the perceived efficacy and/or safety of study treatments. The impact of major protocol deviations on the efficacy and/or safety results will be investigated by assessing the robustness of the study results and conclusions to the choice of analysis set, both including and excluding data potentially affected by major protocol deviations.

Major protocol deviations and any action to be taken regarding the exclusion of subjects or affected data from specific analyses are defined in the Protocol Deviation Specification. A summary of the number and percentage of subjects with major protocol deviation by treatment group and overall and by type of deviation (full analysis set and intent-to-treat analysis set). A by-subject listing of major protocol deviations will be provided.

#### 4.5 Analysis Sets

The **Full Analysis Set** (FAS) consists of all subjects randomized regardless of whether they received study treatment. Subjects will be summarized and analyzed 'as randomized' i.e. by randomized treatment group. If a subject is stratified incorrectly, 'randomized stratum' will be used rather than 'actual stratum'. Summaries of study disposition, protocol deviations and by-subject listings (unless otherwise specified) will be based on the FAS. Efficacy summaries and analyses will be based on the FAS.

The efficacy summaries and analyses will be based on the **intent-to-treat (ITT) analysis set**, which is defined as all randomized subjects who received any amount of study drug. Subjects will be summarized and analyzed 'as randomized' i.e. by randomized treatment group. If a subject is stratified incorrectly, 'randomized stratum' will be used rather than 'actual stratum'.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant

KIN-1901-2001 Statistical Analysis Plan

For the primary and key secondary efficacy endpoints, a sensitivity analysis will be performed on the **per-protocol analysis set** to assess the robustness of the study conclusions to the choice of analysis set. The per-protocol population is defined as all subjects in the ITT **analysis set** who complete the study with no major protocol deviations. A blinded data review will occur prior to the first database lock to decide the subjects being excluded from the per-protocol **analysis set**.

The safety summaries and analyses will be based on the **safety analysis set**. The safety analysis set is defined as all randomized subjects who received any amount of study drug. Subjects will be summarized and analyzed 'as treated' i.e. by actual treatment group.

PK analyses will be based on the **PK analysis set** defined as subjects that receive at least one dose of gimsilumab and have at least 1 evaluable post-dose pharmacokinetic sample.

Upon database release, protocol deviation and analysis set outputs will be produced and will be sent to Kinevant for review. An analysis set classification meeting will be arranged to discuss the outputs and to decide which subjects and/or subject data will be included in the different analysis sets. Such decisions will be made prior to unblinding and will be documented and approved by Kinevant.

A summary of the number and percentage of subjects entering and completing each phase of the study by treatment group and overall for each analysis set (Analysis set: FAS).

A by-subject listing of analysis set details including center, subject identifier, inclusion/exclusion flag for each analysis set and reason for exclusion from an analysis set.

# 4.6 Demographic and Other Baseline Characteristics

Demographic and other baseline characteristics will be summarized by treatment group and for both treatment groups combined (Total) using the ITT analysis set. The summaries provided will include the following.

- Demographic variables:
  - o Age (continuous and categorical (<65 years; ≥65 years))
  - o Sex
  - o Race (American Indian or Alaska Native; Asian; Black or African American; Native Hawaiian or Other Pacific Islander; White; Other; Multiple)
  - o Ethnicity (Hispanic or Latino, Not Hispanic or Latino)
  - o Baseline Height
  - Baseline Weight
  - o Baseline Body Mass Index (BMI)
- Baseline disease characteristics:
  - o Randomization strata (Lung injury/mild ARDS; moderate severe/ARDS)
  - Ventilation status
  - Ventilation type
  - ICU status
  - Oxygenation status
  - Oxygenation type
  - O SpO<sub>2</sub>, FiO<sub>2</sub>, PaO<sub>2</sub>, P/F ratio, S/F ratio
  - o Baseline ferritin, CRP, d-dimer, cardiac troponin I, LDH
  - Baseline Lung Injury Score

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant
KIN-1901-2001 Statistical Analysis Plan

- o Baseline NEWS Total Score
- o Baseline 7-point Ordinal Scale
- o Baseline SOFA Total Score
- $\circ$  Baseline anti-GM-CSF autoantibody concentration (continuous and by categories of <5  $\mu g/mL, \ge 5~\mu g/mL)$
- Days since onset of symptoms

Medical history will be reported by system organ class and preferred term as coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 23.0 or higher.

Age will be reported as calculated in the study database at day of informed consent. BMI will be calculated from baseline height and weight as weight (kg) / height<sup>2</sup> (m<sup>2</sup>).

By-subject listings of demographic data and other baseline characteristics (as summarized above) will be provided.

## 4.7 Prior, Concomitant, and Prohibited Medications and Procedures

Prior and concomitant medications will be summarized by drug class and preferred medication name by treatment group and for both treatment groups combined (Total) using the ITT analysis set . Prior and concomitant medications will be summarized separately, concomitant medications will also be summarized overall and by study period. WHO DDE March 2020 will be used to classify medications.

Medication start and stop dates will be compared to the date of first dose of study drug to allow medications to be classified as either Prior only, both Prior and Concomitant, or Concomitant only. Missing or partial start dates will be imputed as described in <u>Section 4.2.3</u>. Medications starting after the completion/withdrawal date will be listed but will not be classified or summarized.

Medications that start and stop prior to the date of first dose of study drug will be classified as Prior only. If a medication starts before the date of first dose of study drug and stops on or after the date of first dose of study drug, then the medication will be classified as both Prior and Concomitant. Medications will be classified as Concomitant only if they have a start date on or after the date of first dose of study drug.

Use of tocilizumab or any other immunomodulatory biologic (e.g., anti-IL-1, anti-IL-6R, anti-TNF), cell therapies (e.g., mesenchymal stem cells), or small molecules (e.g., JAK inhibitors) is prohibited during the study. Additional prohibited medications may also be defined during blinded data review prior to general study unblinding. The number and percentages of the subjects using such medications will be summarized by treatment groups, and the impact on efficacy and safety will be analyzed by subgroup analyses.

In addition, separate summaries of prior and concomitant steroid use (including the categories 'Any Steroid Use' and 'Any Dexamethasone Use') and other COVID-19 therapies will be provided. Lists of drugs to include in each of these categories will be provided by a medical monitor and the final list will be reviewed and approved prior to general study unblinding.

By-subject listings of prior, concomitant and prohibited medications will be provided. Listings

Effective Date: 30 Jan 19 **Project Document Effective Date**: Date of last signature Related to: SOP-GDO-WW-019 

# 4.8 Efficacy Evaluation

# 4.8.1 Analysis and Data Conventions

# 4.8.1.1 Multi-center Study

The statistical analysis for this multi-center study (with centers quite different in tenns of number of subjects per center) will use the pooled set of subjects across all centers. Center will not be used as a stratification factor or covariate in the statistical analysis models.

## 4.8.1.2 Adjustments for Covariates

The primary efficacy analysis will be adjusted by baseline clinical status (lung injmy/mild ARDS vs moderate/severe ARDS). Baseline clinical status is a randomization factor and the status as repolied from the randomization system will be used for all efficacy analyses.

# 4.8.1.3 Handling of Dropouts or Missing Data

The reason of early study treatment / study discontinuation will be identified, and the percentage of these subjects will be smnmarized by treatment group.

Methodology for multiple imputation and tipping point approaches is described in <u>Section 4.8.1.6</u> and <u>Section 4.8.1.7</u>, respectively.

# 4.8.1.4 Multiple Comparisons/Multiplicity

The one-sided type-I-enor rate (0.025) for the primary efficacy endpoint will be adjusted following the Haybittle-Peto approach with 0.0005 allocated to the interim analysis and 0.0248 allocated to the final analysis.

For the key secondary efficacy endpoints, there is the following serial gate-keeping procedme (also known as sequential conditional testing) addressing the multiplicity and controlling the family-wise one-sided type-I-enor probability to 0.025 (equivalent to two-sided 0.05) for the family of primary and key secondary efficacy endpoints:

- Analysis of the primary efficacy endpoint
   Its null hypothesis is tested on one-sided significance level 0.0248
  - if the null hypothesis cannot be rejected, the entire testing procedure stops here, i.e., null hypotheses for any of the key secondary efficacy endpoints cannot be rejected
  - if the null hypothesis can be rejected, the testing procedure continues with the testing of key secondary efficacy endpoint as described below.
- Analysis of the key secondary efficacy endpoints:
  - A. Survival and no mechanical ventilation on Day 29

Its null hypothesis is tested on one-sided significance level 0.025

- if the null hypothesis is not rejected, the entire testing procedure stops here, i.e., null hypotheses for remaining key secondary efficacy endpoints cannot be rejected
- if the null hypothesis is rejected, the testing procedure continues with the testing of key secondaly efficacy endpoint as described below.
- B. Mechanical ventilation-free days by Day 29

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant KIN-1901-2001

Statistical Analysis Plan

Its null hypothesis is tested on one-sided significance level 0.025

- if the null hypothesis is not rejected, the entire testing procedure stops here, i.e., null hypotheses for the remaining key secondary efficacy endpoint cannot be rejected
- if the null hypothesis is rejected, the testing procedure continues with the testing of key secondaly efficacy endpoint as described below.
- C. Time to hospital discharge by Day 43

Its null hypothesis is tested on one-sided significance level 0.025

- if the null hypothesis is not rejected, the entire testing procedure stops here, i.e., null hypotheses for remaining key secondary efficacy endpoints cannot be rejected
- if the null hypothesis can be rejected, the testing procedure continues with the testing of key secondary efficacy endpoint as described below.

#### 4.8.1.5 Examination of Subgroups

The treatment effect for the primary, key secondaly efficacy endpoints, and the 7-point ordinary scale will be examined for the following subgroups:

- Site
- Clinical status (lung injmy/mild ARDS vs. moderate/severe ARDS)
- Age (<65 yeai·s,65 yeai·s)</li>
- Sex (Male, Female)
- Body weight (by quaiiiles)
- Race (White, African American, additional groups must represent at least 25% of the population if not, will group as 'All Other')
- Ethnicity (Hispanic or Latino, Not Hispanic Latino)
- Invasive ventilator use at baseline (yes, no)
- Baseline invasive ventilator use or severe ARDS at baseline (yes, no)
- Presence of anti-GM-CSF auto antibodies at Screening (<5 μg/mL, 5Lg/mL)
- 7-point ordinal scale status at baseline
- Received Day 8 study dmg (yes, no)
- Prohibited medications use (yes, no) (see <u>Section 4.7</u>)

Prohibited medication use will be aligned to time period of endpoint being summai ized as follows:

- Prohibited medication from Day 1 Day 43 (Mo1iality by Day 43)
- Prohibited medication from Day 1 Day 29 (Smvival and no mechanical ventilation by Day 29, Mechanical ventilation-free days by Day 29)
- Prohibited medication dming the study (Time to hospital discharge, 7-point ordinal scale)

Summaries of the primary, key secondary efficacy vai iables and the WHO 7-point ordinal scale by treatment group and subgroups will be produced.

Homogeneity of the treatment effect across subgroups may be investigated using graphical and analytical methods. An appropriate summaly of the treatment effect (e.g., risk difference, mean difference, hazai·d ratio) and 95% confidence intelvals will be estimated within each subgroup

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

using the methods described for the main analysis for each endpoint. A forest plot showing these estimates and 95% confidence interval within each subgroup and overall will be provided.

# 4.8.1.6 Analysis Methods – Multiple imputation

## General approach

Multiple imputation methods replace each missing primary efficacy endpoint value with a set of m=10 plausible values based on a model predicting values for a missing data point based on available data, i.e., assuming a Missing at Random (MAR) missingness mechanism.

This set of values represents the uncertainty about the correct value to be imputed. These complete datasets (generated by SAS PROC MI) are then analyzed by relevant statistical procedure (e.g., SAS PROC FREQ, SAS PROC LOGISTIC, etc) generating parameter estimates and their standard errors, followed by combining those results from these analyses (by using SAS PROC MIANALYZE).

#### Prediction model

The prediction model attempts to predict a missing endpoint values (e.g, "death by Day 43" or "alive at Day 43" for the binary primary efficacy endpoint) based on available data (variables) that may have an influence on that endpoint.

The proposed prediction model for the binary primary efficacy endpoint is a logistic regression model with the following covariates:

- randomized study treatment: Gimsilumab or placebo
- baseline clinical status: lung injury/mild ARDS or moderate/severe ARDS
- country: USA, etc
- sex: male or female
- age at baseline (continuous covariate)
- body weight at baseline (continuous covariate)
- race (White, African American, additional groups must represent at least 25% of the population if not, will group as 'All Other')
- invasive ventilator use at baseline: no or yes
- anti-GM-CSF auto antibodies at screening: <5 μg/mL or ≥5 μg/mL
- WHO 7-point ordinal scale status at baseline
- National Early Warning Score (NEWS) at baseline
- SpO2 at baseline
- WHO 7-point ordinal scale status at hospital discharge
- NEWS at hospital discharge
- SpO2 at hospital discharge
- second administration of study treatment: yes or no
- administration of prohibited treatments (see Section 4.7) during the study: yes or no

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Algorithm for the multiple imputation of missing values

Within the Bayesian framework, the task of imputing missing values is achieved by drawing random values from the posterior predictive disti·ibution of the missing primary efficacy endpoint data (predicted by the logistic regression prediction model specified above). This posterior predictive disti·ibution is a function of the observed data and regression parameters (or function of regression parameters).

As non-monotone missing pattern may be observed, the fully conditional specification (FCS) method will be used for dealing with arbitiaily non-monotone missing data patterns. The FCS is based on an iterative algorithm; at each iteration and for each vai iable of the prediction model, there is a

- prediction step (P-step): the cmTent (iteration) values of the observed and imputed values are used to derive the predictive distibution of the missing values
- and an imputation step (I-step): updated imputations ai e generated by draws from the predictive disti bution defined by the updated regression model.

When the last vai iable in the sequence (e.g., the primary efficacy endpoint) has been imputed, the algorithm cycles again through each variable, repeating the chain of regression estimation and imputation draw steps. These cycles are repeated and finally there will m=10 draws from the predictive disti-ibution for each missing primary efficacy endpoint value.

Analyzing multiply imputed datasets

Individual statistical analysis (as described in Section 4.8.2 and Section 4.8.3) will be perfo1med for each of the m=IO imputed complete datasets and the results (point estimates and associated standard enors for the study u-eatment effect) will be stored in a single output file.

Estimation and inference for multiply imputed datasets

As a final step, the m=10 estimates and associated standai·d enors will be combined as described below for making statistical inference.

Let Qi and Wi denote the point and vai innce estimates for the study ti eatment effect from the i-th imputed complete data set, i=l, 2,...,m. Then the point estimate for the study ti eatment effect from multiple imputations, Q, is the average of them imputed complete datasets estimates:

$$\bar{Q} = \frac{1}{m} \sum_{i=1}^{m} \hat{Q}_i.$$

Let W denote the average of the m ("within-imputation") variance estimates

$$W=\lim_{m \to \infty} W_{1}$$

and B the estimated ("between-imputation") variance of the point estimates

$$B=\frac{1}{m-1}\operatorname{Im} \stackrel{C}{\mathcal{Q}}_{i-\mathcal{Q}^2}.$$

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant

KIN-1901-2001 Statistical Analysis Plan

Then the total variance V of the multiple imputation estimate  $\mathbb{Q}$  for the study treatment effect is estimated as

$$V = W + (1 + m^{-1}) \cdot B$$
.

Q and Vwill be used for testing null hypotheses stated in <u>Section 4.8.2</u> and <u>Section 4.8.3</u> and constructing two-sided 95% Cis for the study ti eatment effects:

• test statistic

$$t=-\frac{Q}{JV}$$

is approximately disti-ibuted as a I-distribution with degrees of :freedom equal to

$$DFMI = (m-1)(1 + (1+:1) \cdot B)$$

• and the two-sided 95% CI for the study ti eatment effect is calculated as

$$(Q - JV'_{to.975,DFMI}, Q + JV'_{to.975,DFMI}).$$

Where relevant, the exponential function will be used for ti ansfonning point estimates and CI limits from the log scale to the original scale.

# 4.8.1.7 Analysis Methods - Tipping point analysis

Graphical displays, based on the "tipping-point" analysis intioduced by <u>Yan 2009</u> and not requiring the MAR assumption, will be used to visualize the results of a two-dimensional set of sensitivity analyses using different imputations for missing binaiy endpoint values (e.g., either "death by Day 43" or "alive at Day 43" for the primaiy efficacy endpoint) for compairison of the two study t:I'eatments. All possible combinations of imputations of missing binaiy endpoint values in the gimsilumab and placebo group will be evaluated by the statistical method described in Section 4.8.2 and Section 4.8.3, with study tireatment as the only factor.

<u>Figure 4-1</u> below is an example graphic taken from Campbell 2011 with 8 missing endpoint values in the "Treatment Group" (one can impute Oto 8 successes) and 11 missing endpoint values in the "Cont:I'ol group" (one can impute O to 11 successes), leading to a mati·ix of 108 (= 9 times 12) combinations to be tested. For the example displayed in <u>Figure 4-1</u>, 10 combinations close to the upper left upper comer "worst case" (all missing values in the "Cont:I'ol Group" were imputed as successes and all missing value in the "Treatment Group" were imputed as failures) did not lead to a significant test result (rejection of the null hypothesis).

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Figure 4-1 Example for a tipping point analysis summary display



"Enhanced tipping-point displays" (<u>Liublinska 2014</u>) will be provided as compact summaries of conclusions drawn from different alternative assumptions.

## 4.8.1.8 Analysis Methods - Final analysis following adaptive sample size increase

"Successes" In Missing in Treatment Group

If the sample size has been increased at interim analysis 2 (see <u>Section 5.2.5</u>), then the final analysis of the primary efficacy endpoint (moliality by Day 43) and key secondary endpoints will be perfolmed by using a weighted average of the two one-sided test statistics Z1 and Z2 based on data from subjects in stage 1 and stage 2 sepai ately, respectively.

The test statistic *ZcHw* (maintaining the type-l-eITor probability restricted to one-sided 0.0248 (primary endpoint) or 0.025 (key secondaly endpoints) per <u>Cui/Hung/Wang 1999</u>) for the final analysis will be

$$ZcHw = w_1 \cdot Z_1 + w_2 \cdot Z_2$$

and the pre-specified weights are

 $w_1 = \underline{ffe}$  with  $n_1$  denoting the number of subjects in the FAS for stage 1

 $w_2 = \int_{-\infty}^{\infty} \frac{1}{n}$  where 270 -  $n_1$  represents the number of subjects in the FAS for stage 2.

## 4.8.1.9 Analysis Methods - Continuous vai iables

All continuous outcomes will be sUffilnai ized using descriptive statistics by treatment group and visit. For each outcome only planned visits as detailed in the schedule of assessments (Appendix 7.1) will be summarized.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant KIN-1901-2001

Statistical Analysis Plan

# 4.8.1.10 Analysis methods - Count variables

For number of event-free days (mechanical ventilation free days, ICU-free days) the median, 1<sup>st</sup> qualiile and 3<sup>rd</sup> qualiile will be presented by treatment. A Wilcoxon rank sum test will be used to evaluate the difference between treatment groups.

# 4.8.1.11 Analysis methods - Categorical vai iables

For binaly endpoints the number and propoliion in each treatment group will be presented along with the common risk difference with 95% CI (gimsilumab - placebo) as estimated using the Mantel-Haenszel method. Baseline clinical status will be used as stratification factor. A Cochran-Mantel-Haenszel (CMH) test may be used to test for a treatment effect.

Binaiy primaiy and key secondaiy endpoints will also be evaluated with common risk difference obtained from logistic regression (following <u>Ge et al 2011)</u> with covariates study treatment and baseline clinical status

Other categorical outcomes will be evaluated using CMH tests stratified for baseline clinical status.

# 4.8.1.12 Analysis Methods - Time to event variables

Time to event analyses will be perfonned using Kaplan-Meier method and a log-rank test stratified by baseline clinical status will be used to evaluate the treatment effect (gimsilumab vs. placebo). The total number of subjects with an event, the total number censored, reasons for censoring, and Kaplan-Meier estimates with associated 95% Cis for survival probabilities at Days 15, 29, 43, 85, 169 as well as 25<sup>th</sup> percentile, median, and 75% percentile (if available) survival time and 95% Cis will be presented bytreatment group. Survival plots or cumulative incidence plots as specified for each time to event endpoint will be presented by treatment and by randomization strata (baseline clinical status) and treatment. If one of the baseline clinical status categories have fewer than 10 events overall, Kaplan-Meier estimates will only be presented overall.

A propoliional hazard model stratified by baseline clinical status (if there are sufficient events in each stratum) will be used to estimate the hazai d ratio and associated 95% CI of gimsilumab vs. placebo.

#### 4.8.1.13 Analysis Methods - Multi-state competing risks models

For time to hospital discharge and time to clinical improvement a supplementary analysis using a multi-stat competing risks model will be perfo1med (Beyersmann, Allignol, Schumacher 2012).

# Multi-state competing risks model

For each subject, a multi-state stochastic process (Xd)tkO is considered where Xd denotes the state a subject is in at the end of day d, 1 :S d '.S 43 (43 is the final day of the planned observation period Three states are defined as follows:

[Baseline] baseline state

[Improvement] improvement state (assumed as an absorbing state as further transitions ai e not considered here)

[Death] death state (absorbing state)

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant

KIN-1901-2001 Statistical Analysis Plan

All subjects stail in the initial state [Baseline] at time of randomization, d=0, i.e.,  $x_0 =$  [Baseline]. If subject recovers but dies (aftelwai·ds) on the same day d, then that subject's state  $x_d$  will be set to  $x_d =$  [Death].

States and possible transitions between states are illustrated by Figure 1 below.

Figure 1 Competing risks model



A transition probability from state [Baseline] at day  $_{\sigma}$  (0  $_{\sigma}$  42) to state  $_{[m]}$  at day  $_{\sigma}$   $_{\sigma}$  43, is defined as:

P[Baseline)[m](d, e) = P(Xe = [m]IXd = [Baseline])

Subjects stay in state [Baseline] as long as none of the competing events have occuned; the competing risks process moves out of the [Baseline] state at day *TD*, defined as

$$TD = \min\{d > OIXd^* \text{ [Baseline]}\}\$$

and is called the transition day; state Xm is the type of transition.

The competing risks process is subject to right-censoring (assumed to be independent of the transition processes) when a subject's follow-up was terminated while the subject was still in state [Baseline]:

- either prematurely prior to the end of Day 43
- or when reaching the planned end of observation period at end of Day 43.

The hazai of functions for transitions from state [Baseline] to state [Improvement] or to state [Death], respectively, ai e assumed to detennine the stochastic behavior of the competing risks process; these hazai of functions differ bystudy treatment group.

The transition-specific cumulative incidence functions over the 43 days observation period are defined as Pk, c(D :::; d, Xv = [m]), where [m] can be state [Improvement] or state [Death], k denotes the stratum and c the study treatment (gimsilumab or placebo) will be derived from non-parametric Nelson-Aalen estimators for cumulative hazai d functions.

## Stratified transition-specific proportional hazards models

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant
KIN-1901-2001
Statistical Analysis Plan

The transition-specific proportional hazards model stratified for factors used in the randomization and its assumptions are illustrated by:

 $h_{[\text{Baseline}],[m]}(d, x_{jk}, \beta_{[\text{Baseline}],[m]}) = h_{[\text{Baseline}],[m];0k}(d) \cdot \exp(x_{jk} \cdot \beta_{[\text{Baseline}],[m]})$ 

 $h_{[Baseline],[m]}(.)$  transition-specific hazard functions as a function of days (relative to date of randomization), the subject's stratum and study treatment (gimsilumab or placebo), and unknown hazard ratio

 $h_{[\text{Baseline}],[m];0k}(d)$  unspecified transition-specific hazard function for placebo subjects in stratum

k at day d; transition-specific hazard functions for placebo are allowed to vary

across strata without any restrictions

 $x_{jk}$  study treatment indicator for subject j in stratum k, coded as 0 for placebo, 1 for

gimsilumab

 $h_{[\text{Baseline}],[m]}$ : vector of unknown transition-specific log hazard ratios for study treatment;

assumed to be common across strata, allowed to differ by transition.

Estimation of transition-specific hazard ratios will be performed by maximizing partial likelihood functions; two-sided 95% confidence intervals will be provided.

4.8.1.14 By-subject listings

All derived efficacy endpoints and the raw data points used to derive them will be listed by subject.

# 4.8.2 Analysis of the Primary Efficacy Endpoint

<u>Clinical question of interest:</u> Does gimsilumab reduce mortality (up to Day 43) in subjects with lung injury or ARDS secondary to COVID-19 in comparison to placebo?

<u>Intercurrent events</u> (may occur between randomization and Day 43), not mutually exclusive:

- IE1: subject's withdrawal from the study prior to Day 43
- IE2: subject lost to follow-up prior to Day 43
- IE3: subject did not receive any dose of study treatment

## Attributes of Estimand 1 (following a treatment policy strategy)

- A. Patient population: as defined by protocol eligibility criteria and treated
- B. Treatment conditions:
  - condition of interest: randomized to gimsilumab and treated
  - alternative/control condition: randomized to placebo and treated
- C. Endpoint: subject's death by Day 43
- D. <u>Population-level summary</u>: estimated incidence probability for death up to Day 43 (in each treatment group separately)

Main estimator for Estimand 1: common mortality risk difference (for death up to Day 43) across both strata defined by baseline clinical status used in the stratified randomization

• Intercurrent events IE1 and IE2 will be disregarded for the inclusion of subjects in the statistical analysis, IE3 restricts the inclusion of subjects to those who received at least one dose of study treatment. Hence, the main estimator for Estimand 1 will be based on the ITT analysis set.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant
KIN-1901-2001 Statistical Analysis Plan

• For subjects with missing primary endpoint data resulting from !El and IE2, a multiple imputation approach (details see <a href="Section 4.8.1.6">Section 4.8.1.6</a>) assuming MAR will be used. The set of complete (imputed) datasets will be analyzed as 2x2 frequency tables strntified by baseline clinical status obtaining Mantel-Haenszel common risk difference estimates and respective standard enors for those datasets. These results will then appropriately combined (see <a href="Section 4.8.1.6">Section 4.8.1.6</a>) to obtain point estimate and CI for the common risk difference as well as for a one-sided p-value for testing the null hypothesis of a common moliality risk difference 0.

<u>Sensitivity estimators for Estimand 1</u> (also based on the ITT analysis set):

- Two-dimensional tipping point analysis vaiying the missing primary endpoint data in the two study treatment aims (see <u>Section 4.8.1.7</u>) not assuming MAR
- Common moliality risk difference (for death up to Day 43) obtained from logistic regression (following <u>Ge et al 2011)</u> with covai intes study treatment and baseline clinical status (and multiple imputation approach described in <u>Section 4.8.1.6</u> assuming MAR).

<u>Supplementary analysis</u>: Overall smyival will be analyzed using time to event methods as described in <u>Section 4.8.1.12</u>. Time to death is defined as the time from randomization to death in days (*date of death - randomization date* + 1). Subjects without a recorded death will be censored at their last date known alive (completion date if they were followed through Day 169 or at their early discontinuation date if they withdrew early or at their date of last assessment if they ai e alive and ongoing in study at time of analysis; *last date known alive - randomization date* +J).

Eugpl fuantluly5 Secondaiy) analysis: Main estimator analysis will be repeated for moliality by

## Attributes of Estimand 2 (following a composite policy strategy)

- A. Patient population: as defined by protocol eligibility criteria and treated
- B. Treatment conditions:
  - condition of interest: randomized to gimsilumab and treated
  - alternative/control condition: randomized to placebo and treated
- C. <u>Endpoint:</u> subject's death by Day 43 or subject withdrawn from the study prior to Day 43 or subject got lost to follow-up prior to Day 43
- D. <u>Population-level summaiy</u>: estimated incidence probability for death by Day 43 or study withdrawal prior to Day 43 or lost to follow-up prior to Day 43 (in each treatment group sepai ately)

<u>Main estimator for Estimand 2</u>: common risk difference across both strata defined by baseline clinical status used in the stratified randomization

• !El and IE2 are pait of the composite endpoint, so these two!Es will be disregarded for the inclusion of subjects in the statistical analysis, IE3 restricts the inclusion of subjects to those who received at least one dose of study treatment. Hence, the main estimator for Estimand 2 will be based on the ITT analysis set and none of the subjects have a missing composite endpoint value.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Sensitivity estimators for Estimand 2 (also based on the ITT analysis set):

• Common risk difference obtained from logistic regression (following <u>Ge et al 2011)</u> with covariates study treatment and baseline clinical status

<u>Supplementary analysis:</u> time to death or withdrawal or lost to follow-up will be analyzed using time to event methods as described in <u>Section 4.8.1.12</u>. Time to death or withdrawal is defined as the time from randomization to death or withdrawal in days (*date of death/withdrawal* -  $randomization \ date + 1$ ). Subjects without a recorded death or withdrawal will be censored at their last date known alive in the study (completion date if they were followed through Day 169 or othelwise at their date of last assessment; *last date known alive in the study* -  $randomization \ date + 1$ ).

# 4.8.3 Key Secondary Efficacy Analysis

4.8.3.1 Survival and no mechanical ventilation on Day 29

<u>Clinical question of interest:</u> Does gimsilumab reduce mechanical ventilation on Day 29 and m01iality up to Day 29 in subjects with lung injury or ARDS secondary to COVID-19 m comparison to placebo?

<u>futercmTent events</u> (may occur between randomization and Day 29), not mutually exclusive:

- IEl: subject's discharge from the hospital prior to Day 29
- IE2: subject's withdrawal from the study prior to Day 29
- IE3: subject lost to follow-up prior to Day 29
- IE4: subject did not receive any dose of study treatment

#### Attributes of Estimand 2-1 (following a composite policy strategy)

- A. Patient population: as defined by protocol eligibility criteria and treated
- B. Treatment conditions:
  - condition of interest: randomized to gimsilumab and treated
  - alternative/control condition: randomized to placebo and treated
- C. <u>Endpoint:</u> subject is alive and not on mechanical ventilation on Day 29 or discharged prior to Day29
- D. <u>Population-level summaiy</u>: estimated probability of being alive and not on mechanical ventilation on Day 29 (in each treatment group separately)

<u>Main estimator for Estimand 2-1</u>: common risk difference across both strata defined by baseline clinical status used in the stratified randomization

- futercmTent events IEl is included in the endpoint definition: subjects dischai ged alive prior to Day 29 (IEl) are considered successes for this endpoint as it is assumed that mechanical ventilation is no longer necessaiy for subjects who have been discharged from the hospital.
- futercmTent events IE2 and IE3 will be disregarded for the inclusion of subjects in the statistical analysis; IE4 restricts the inclusion of subjects to those who received at least one dose of study treatment. Hence, the main estimator for Estimand 2-1 will be based on the ITT analysis set.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant
KIN-1901-2001 Statistical Analysis Plan

• For subjects with missing primary endpoint data resulting from IE2 and IE3, a multiple imputation approach (details see Section 4.8.1.6) assuming MAR will be used. The set of complete (imputed) datasets will be analyzed as 2x2 frequency tables strntified by baseline clinical status obtaining Mantel-Haenszel common risk difference estimates and respective standard enors for those datasets. These results will then appropriately combined (see Section 4.8.1.6) to obtain point estimate and confidence interval (CI) for the common risk difference as well as for a one-sided p-value for testing the null hypothesis of a common risk difference 0.

### Sensitivity estimators for Estimand 2-1:

- Two-dimensional tipping point analysis vaiying the missing primary endpoint data in the two study treatment aims (see <u>Section 4.8.1.7</u>)
- Common response probability difference obtained from logistic regression (following Ge et al 2011) with covai intesting study ti eatment and baseline clinical status (and multiple imputation approach described in Section 4.8.1.6).

<u>Supplementary</u> (Secondary) analysis: Main estimator analysis will be repeated for probability of being alive and not on mechanical ventilation on Days 15, 22, and 43.

4.8.3.2 Mechanical ventilation-free days by Day 29

<u>Clinical question of interest:</u> Does gimsilumab increase the number of mechanical ventilation-free days up to Day 29 in subjects with lung injmy or ARDS secondary to COVID-19 in comparison to placebo?

<u>Intercmrent events</u> (may occm between randomization and Day 29), not mutually exclusive:

- !El: subject's death prior to Day 29
- IE2: subject discharge (alive) from the hospital prior to Day 29
- IE3: subject's withdrawal from the study prior to Day 29 and prior to hospital discharge
- IE4: subject did not receive any dose of study ti eatment

#### Attributes of Estimand 2-2 (following a composite policy strategy)

- A. Patient population: as defined by protocol eligibility criteria and ti-eated
- B. Treatment conditions:
  - condition of interest: randomized to gimsilumab and ti-eated
  - alternative/conti·ol condition: randomized to placebo and ti·eated
- C. Endpoint: subject's number of mechanical ventilation-free days by Day 29
- D. <u>Population-level summaiy:</u> median number of days not on mechanical ventilation by Day 29 (in each ti-eatment group separately)

<u>Main estimator for Estimand 2-2</u>: difference of medians for number of days not on mechanical ventilation by Day 29.

- Mechanical ventilation status (yes/no) will be assessed daily while subjects remain hospitalized up to and including their date of dischaige.
- For a subject who died prior to Day 29 (IEI), the number of mechanical ventilation-free days up to Day 29 will be set to 0.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant
KIN-1901-2001
Statistical Analysis Plan

- For a subject alive at Day 29 and hospitalized at least up to Day 29, the number of mechanical ventilation-free days up to Day 29 is the sum of days with mechanical ventilation status of 'no' from Day 1 through Day 29.
- For a subject discharged from hospital alive prior to study day 29 (IE2), the number of mechanical ventilation-free days up to Day 29 is the sum of
  - (1) the number of days with mechanical ventilation status of 'no' from Day 1 to date of hospital discharge and
  - (2) the number of days from their date of discharge through their Day 29 visit (Day 29 visit date date of discharge), assuming that a subject is not mechanically ventilated after hospital discharge.
- For a subject who withdrew from the study prior to Day 29 and prior hospital discharge (IE3), the number for mechanical ventilation-free days will be the sum of days with mechanical ventilation status of 'no' from Day 1 through the day of study withdrawal.
- Intercurrent event IE3 will be disregarded for the inclusion of subjects in the statistical analysis; IE4 restricts the inclusion of subjects to those who received at least one dose of study treatment. Hence, the main estimator for Estimand 2-2 will be based on the ITT analysis set.

The number of mechanical ventilation-free days will be analyzed by a Wilcoxon rank sum test stratified by baseline clinical status to obtain a one-sided p-value for testing the null hypothesis of equal or more favorable distribution for placebo compared to gimsilumab.

<u>Supplementary (Secondary) analyses</u>: Main estimator analysis will be repeated for mechanical ventilation-free days by Days 15, 22, and 43.

# 4.8.3.3 Time to hospital discharge

<u>Clinical question of interest</u>: Does treatment with gimsilumab result in a shorter overall duration of hospitalization in subjects with lung injury or ARDS secondary to COVID-19 in comparison to placebo?

#### Intercurrent events:

- IE1: subject's death prior to hospital discharge
- IE2: subject's withdrawal from the study prior to hospital discharge
- IE3: subject did not receive any dose of study treatment

# **Attributes of Estimand 2-3 (following a composite policy strategy)**

- A. Patient population: as defined by protocol eligibility criteria and treated
- B. Treatment conditions:
  - condition of interest: randomized to gimsilumab and treated
  - alternative/control condition: randomized to placebo and treated
- C. Endpoint: subject's time to hospital discharge
- D. <u>Population-level summary</u>: median time to hospital discharge (in each treatment group separately)

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant KIN-1901-2001

Statistical Analysis Plan

<u>Main estimator for Estimand 2-3</u>: hazard ratio across combined strnta defined by baseline clinical status used in the stratified randomization (see <u>Section 4.8.1.12</u> for details)

- Time to hospital discharge is the time in the hospital after randomization in days (Table 4-
- **i** that case that a subject is still hospitalized at time of analysis they will be censored at their date of last assessment in the data cut.
- Subjects who die before leaving the hospital (IEI) will be considered failures (did not achieve hospital discharge) and will continue to contribute to the risk pool through the end of the analysis period, that is they will be censored at the date of data cut.
- ill the case that a subject withdraws from the study before leaving the hospital (IE3), they will be censored at their discontinuation date, respectively.
- IE3 restricts the inclusion of subjects to those who received at least one dose of study treatment. Hence, the main estimator for Estimand 2-3will be based on the ITT analysis set.

<u>Sensitivity estimator</u>: Analyses for main estimator will be repeated using a modified definition of time to hospital discharge where subjects who died (IEI) are censored at time of death. <u>Table 4-2</u> provides endpoint derivation details.

Table 4-2: Time to hospital discharge definitions

| Carbinata status at time of | Main estimator * | | Sensitivity estimator* | |
|---|---|---|---|---|
| Subjects status at time of analysis: | Event date | Censored (yes/no) | Event date | Censored (yes/no) |
| Alive, discharged from hospital | Date of discharge | No | Date of discharge | No |
| Alive, still hospitalized | Date oflast assessment | Yes | Date oflast assessment | Yes |
| Early withdrawal from study<br>before discharged from hospital<br>(IE2) | Date of early withdrawal | Yes | Date of early<br>withdrawal | Yes |
| Lost to follow-up before discharged from hospital (IE3) | Date oflast assessment | Yes | Date oflast assessment | Yes |
| Died (IEI) | Date of data cut | Yes | Date of death | Yes |
| *Time to hospital dischar e will be repolted in days and defined as event date - randomization date + 1. | | | | |

<u>Supplementaly analysis</u>: A multi-state competing risks model will be perfolmed as described in <u>Section 4.8.1.13</u> replacing the improvement state by hospital discharge.

## 4.8.4 Other Secondary and Exploratory Efficacy Analyses

Other secondary and exploratoly endpoints will be analyzed according to the type of endpoint as described below. If data are sparse for any of the exploratory endpoints, summaries may be limited to descriptive statistics of available data or listings only as appropriate.

#### ICU-free days by Days 15, 22, 29 and 43

This endpoint will be defined and analyzed similarly to mechanical ventilation-free days (Section 4.8.3.2). ICU status (yes/no) will be assessed daily while subjects remain hospitalized up to and

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 
Statistical Analysis Plan

including their date of discharge. For subjects who are alive at the time of analysis and remain hospitalized the number of days with ICU status of 'no' from day of first dose through their Day 15 (22/29/43) visit will be summed. For subjects who are alive at time of analysis visit but have been discharged prior to study Day 15 (22/29/43), the total number of ICU-free days will be the sum of (1) the number of days with ICU status of 'no' will be summed through their date of discharge and (2) the number of days from their date of discharge through their Day 15 (22/29/43) visit (Day 15 (22/29/43) visit date – date of discharge). For subjects who died at time of analysis the number of ICU-free days will be set to 0. For subjects with missing data due to early study withdrawal prior to hospital discharge, the number for ICU-free days will be the sum of days with ICU status of 'no' from Day 1 through the day of study withdrawal. The median, 1<sup>st</sup> quartile, and 3<sup>rd</sup> quartile of the number of ICU-free days will be presented for each treatment group. A Wilcoxon rank sum test will be used to test the null hypothesis that there is no difference in number of ICU-free days between gimsilumab and placebo (Section 4.8.1.10).

### Incidence of mechanical ventilation use Overall and by Days 15, 22, 29 and 43

This endpoint will be evaluated for all subjects, no matter if the subject was on or not on a mechanical ventilator at the time of the randomization. Mechanical ventilation use by Day 15 (22/29/43) will be defined as 'Yes' if subject is alive and was on mechanical ventilation on or prior to Day 15 (22/29/43). As ventilation status is only collected while subject remains in the hospital, subjects who were discharged before Day 15 (22/29/43) and are still alive will be considered not be on mechanical ventilation. Subjects missing data due to death, early study withdrawal, or lost to follow-up prior to Day 15 (22/29/43) will be considered 'on mechanical ventilation'.

The number and percentage of subjects achieving this endpoint will be summarized by treatment group. In addition, the common mechanical ventilation use risk difference across both strata defined by baseline clinical status used in the stratified randomization with 95% CI will be reported.

Among subjects with mechanical ventilation, median, 25<sup>th</sup> percentile and 75<sup>th</sup> percentile (with 95% confidence intervals) estimated using Kaplan-Meier method will be used to summarize duration of mechanical ventilation and time to first mechanical ventilation. Duration of mechanical ventilation will be summarized for subjects on mechanical ventilation separately for ventilation starting at baseline and ventilation starting post-baseline. Duration of mechanical ventilation will only be derived for subjects who are removed from ventilation (end date of ventilation – start date of ventilation + 1) or who died while still on ventilation (date of death – start date of ventilation + 1).

Time to first mechanical ventilation will be summarized only for subjects starting mechanical ventilation post-baseline and is defined as time from randomization to first date of mechanical ventilation for subjects who started ventilation post-baseline.

#### Incidence of ICU use by Days 15, 22, 29 and 43

Incidence of ICU use will be defined and analyzed similarly to incidence of mechanical ventilation use using the daily assessments of ICU status taken while subjects are hospitalized.

#### NEWS and SOFA scores

Standard descriptive statistics (mean, standard deviation, median, minimum, maximum) will be used to summarize each of these scores by treatment group and visit. NEWS and SOFA (total and component scores) scores will be assessed daily while subject is hospitalized. Plots of mean score

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Statistical Analysis Plan

(with standard error bars) by treatment group over time may be produced. SOFA component scores are respiratory score, cardiovascular score, liver score, renal score, coagulation score, and neurologic score.

Figure 4-2: National Early Warning Score (NEWS)

| PHYSIOLOGICAL<br>PARAMETERS | 3 | 2 | 1 1 | 0 | 1 | 2 | 3 |
|---|---|---|---|---|---|---|---|
| Respiration Rate | ≤8 | | 9 - 11 | 12 - 20 | | 21 - 24 | ≥25 |
| Oxygen<br>Saturations | ≤91 | 92 - 93 | 94 - 95 | ≥96 | | | |
| Any Supplemental<br>Oxygen | | Yes | | No | | | |
| Temperature | ≤35.0 | | 35.1 - 36.0 | 36.1 - 38.0 | 38.1 - 39.0 | ≥39.1 | |
| Systolic BP | ≤90 | 91 - 100 | 101 - 110 | 111 - 219 | | | ≥220 |
| Heart Rate | ≤40 | | 41 - 50 | 51 - 90 | 91 - 110 | 111 - 130 | ≥131 |
| Level of<br>Consciousness | | | | А | | | V, P, or U |

#### 7-point ordinal scale

The 7-point ordinal scale is as follows:

- 1. Not hospitalized, no limitations on activities;
- 2. Not hospitalized, limitation on activities;
- 3. Hospitalized, not requiring supplemental oxygen;
- 4. Hospitalized, requiring supplemental oxygen;
- 5. Hospitalized, on non-invasive ventilation or high-flow oxygen devices;
- 6. Hospitalized, on invasive mechanical ventilation or ECMO;
- 7. Death.

The 7-point ordinal scale represents the worst status on the day prior to the visit, that is, assessment collected on Day 2 is reported for Baseline (Day 1), assessment collected on Day 3 is reported for Day 2, etc. As data is not expected to be reported the day after a subject's death, hence a score of 7/"Death" will be imputed on the date of death for analysis purposes. No visit windowing will be applied. For example, for subjects who were discharged from the hospital prior to Day 15 their results from follow-up visit Day 15 are reported on Day 14 regardless of actual study day result was recorded for.

The percentage of subjects reporting each severity rating (1-7) of the 7-point ordinal scale and shift from baseline category will be reported for all study days (Daily while hospitalized and then on Days 15, 22, 29, 35, 43, 85, and 169/EoS). The percentage of subjects with change in ordinal scale at these time points will also be summarized for each of the following:

- 1-point improvement from baseline
- 2-point improvement from baseline

TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

Statistical Analysis Plan

- 3-point improvement from baseline
- ≥4-point improvement from baseline
- No change from baseline
- 1-point worsening from baseline
- 2-point worsening from baseline
- 3-point worsening from baseline
- 4-point worsening from baseline

Shift tables comparing score at baseline to last assessment available for each subject will be created overall and by subgroup.

Stacked bar plots by treatment group and visit (Baseline, Days 7, 14, 21, 28, 35, 42, 84 and 168) will be produced for 7-point scale results and change from baseline (excluding baseline visit).

#### Time to first clinical improvement

Time to first clinical improvement is defined as the earliest of (1) first time the 7-point ordinal scale shows a 2-point decrease from the baseline score or (2) discharge from the hospital (date of first clinical improvement - first dose date + 1) for subjects who achieved clinical improvement and are still alive at time of analysis. Subjects who did not achieve a 2-point reduction and are still alive at time of analysis will be censored at their date of last assessment. Subjects who died will be treated as failures (did not achieve clinical improvement) and will continue to contribute to the risk pool through the end of the analysis period, that is they will be censored at the date of data cut. Kaplan-Meier method will be used to estimate the median time to clinical improvement (Section 4.8.1.12) and a cumulative incidence plot will be provided.

<u>Supplementary analysis:</u> A multi-state competing risks model will be performed as described in <u>Section 4.8.1.13</u> replacing the improvement state by first clinical improvement (earliest of 2-point decrease from baseline in 7-point ordinal scale score or hospital discharge).

#### Oxygen-free days during hospitalization

Oxygen use status (yes/no) will be assessed daily while subjects remain hospitalized up to and including their date of discharge. For subjects who are alive at the time of analysis and remain hospitalized the number of days with oxygen status of 'no' from day of randomization through their Day 15 (22/29/43) visit will be summed. For subjects who died at time of analysis the number of Oxygen-free days during the hospitalization will be set to 0. Descriptive statistics by treatment group and a treatment group comparison of number of days not oxygen by Day 15 (22/29/43) using a Wilcoxon rank sum test as described in Section 4.8.1.10.

#### Incidence of ECMO use and duration

The number and percentage of subjects using ECMO while on study will be summarized by treatment. For subjects who used ECMO the duration in days will be summarized using descriptive statistics.

<u>Change from baseline in respiratory outcomes, select laboratory test results, COVID-19 viral load, and LVEF</u>

Respiratory outcomes include the secondary endpoint SpO<sub>2</sub>/FiO<sub>2</sub> and the exploratory endpoints lung injury score (LIS), and PaO<sub>2</sub>/FiO<sub>2</sub>. Laboratory test endpoints include D-dimer, cardiac troponin I, lactate dehydrogenase (LDH), ferritin, procalcitonin, and C-reactive protein (CRP) as

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant

KIN-1901-2001 Statistical Analysis Plan

secondaly endpoints. COVID-19 viral load as measured by quantitative PCR is a secondaiy endpoint, and LVEF is an optional cardiovascular assessment and exploratoly endpoint.

Standard descriptive statistics (mean, standai deviation, median, minimum, maximum) will be used to summarize each outcome and it's change from baseline bytreatment group and visit. Only scheduled visits as described in the schedule of assessments (Appendix 7.1) will be included for each endpoint.

For select endpoints, mean (with standard enor bars) results and change from baseline may be plotted over time by treatment group.

Exploratoly endpoints (LIS, PaO2/FiO2, LVEF) will only be summarized by visit if at least 20% of subjects have at least one non-missing assessment, othelwise only by-subject listings will be provided for these endpoints. Chest radiographic results will be provided in a by-subject listing.

### 4.9 Safety Evaluation

All safety summaries and analyses will be based upon the safety analysis set as defined in <u>Section 4.5</u>. Safety analyses summarized by study period will be analyzed separately for each of the following periods as defined in <u>Section 4.2.1</u>:

- Overall
- Treatment Period (Day 1 -Day 15)
- Follow-up Period 1 (Day 16-Day 43)
- Follow-up Period 2 (Day 44 +)
- Overall-Hospitalized (Day 1 through DoD)
- Overall After Discharge (DoD +)

Note: only subjects who were on study in a given period will be included in the analysis for that period (e.g. if a subject withdraws from study or dies before Day 43 they will contribute to the denominator for summaries in the Overall, Treatment Period, and Follow-up Period 1 periods, but not in summaries of Follow-up Period 2).

#### 4.9.1 Extent of Exposure

The number and percent of subjects that were dosed at each planned dose (Day 1 and Day 8) will be presented by treatment group. The number and percent of dose inteln1ptions will also be summarized by treatment group. The daily dose at days 1 and 8 and cumulative dose will be presented by treatment group using descriptive statistics. A by-subject listing of exposure data will be provided.

#### 4.9.2 Adverse Events

Adverse events will be coded using the Medical Dictionaiy for Regulatory Activities (MedDRA) Version 23.0 or higher.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant

KIN-1901-2001 Statistical Analysis Plan

Treatment-emergent adverse events will be tabulated and are defined as those adverse events that either stail or worsen in severity on or after the date/time of first dose of study treatment and through the end of safety follow-up period.

Where dates are missing or paiiially missing, adverse events will be classified as treatment emergent and into study periods using imputed dates as described in <u>Section 4.2.3</u>.

An overall summaiy table of treatment-emergent AEs (TEAEs) will be provided with the number and percentage of patients (incidence) repoliting an event along with the total number of events presented for the following categories:

- All TEAEs (all grades and grades 3-5)
- Study dmg-related TEAEs (all grades and grades 3-5)
- Serious TEAEs
- Study dmg-related SAEs
- Fatal TEAEs
- TEAEs leading to study diug discontinuation
- Each AESI (see Section 4.9.2.2)

### 4.9.2.1 AE Summaries bysystem organ class (SOC) and prefened te1m (PT)

The incidence and total number of events for the following will be sUillllai ized by SOC and PT:

- All TEAEs
- Study dmg-related TEAEs
- TEAEs by maximum severity
- Study dmg-related TEAEs by maximum severity
- Grade 3 or higher TEAEs
- Study dmg-related grade 3 or higher TEAEs
- Serious TEAEs
- Dmg-related SAEs
- Fatal Serious TEAEs
- TEAEs leading to study diug discontinuation
- Each AESI (see Section 4.9.2.2)

Adverse events will be summarized by treatment overall and by study period. Adverse event summaries will be ordered by decreasing frequency for SOC, and PT within SOC, in the gimsilumab treatment group, and then similaily by decreasing frequency in the placebo treatment group, and then alphabetically for SOC, and PT within SOC.

For each subject and each adverse event, the worst severity recorded will be attributed and used in the by-severity summaries. Similarly, the worst causality (most related to treatment) will be attributed and used in the by-causality summaries. If severity or causality is missing, the worst case will be assumed.

### 4.9.2.2 AE of Special Interest (AESI)

AESI will be defined using standard MedDRA queries (SMQ). See <u>Appendix 7.3</u> for a complete list of terms. The following TEAEs are of special interest:

| Adverse Event of Special Interest | Include all terms (Narrow and Broad) from SMQs |
|---|---|
| Clinically severe or life-threatening onset of new infections (besides COVID-19) | Infective Pneumonia Opportunistic Infections Note: include only events with severity of 'Severe' or 'Life-threatening', exclude PTs 'Coronavirus infection' 'Coronavirus test positive' |
| Neutropenia, Thrombocytopenia, and Leukopenia | Hematopoietic Cytopenia |
| Injection related reactions | Hypersensitivity Reaction Drug Reaction Anaphylactic reaction |
| Transaminitis | Hepatic Disorders- Drug related hepatic disorder |
| Pulmonary alveolar proteinosis | Interstitial Lung Disease |

### 4.9.2.3 Adverse event listings

By-subject listings of all adverse events (including non-treatment-emergent events) will be provided. This listing will be presented by treatment group and will include center, subject identifier, age, sex, race, adverse event (SOC, PT, and verbatim term), date of onset, date of resolution, study period, hospitalization status, duration, severity, seriousness, action taken, outcome and causality. The following listings will be provided:

- All adverse events
- All drug-related adverse events
- All grade 3-5 adverse events
- All serious adverse events
- All fatal adverse events
- All adverse events leading to discontinuation of study treatment
- All adverse events of special interest

#### 4.9.3 Clinical Laboratory Evaluation

The following laboratory parameters will be summarized by treatment group and visit for each study period using appropriate descriptive statistics.

| Hematology | Chemistry | Coagulation |
|------------|-----------|------------------|
| Hemoglobin | BUN | Prothrombin time |

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant

KIN-1901-2001 Statistical Analysis Plan

Activated paliial Creatinine

Hematocrit thromboplastin time (aPTT)

Fibrinogen **Platelets** Glucose **Urinalysis** Red blood cells Sodium Glucose White bloods cells Potassium Neutrophils Chloride Protein Lymphocytes Total CO2 Ketones

Monocytes Calcium Specific gravity

Alanine aminotransferase Eosinophils рН

(ALT

Aspaiiate aminotransferase Basophils Blood

(AST) Albumin **Nitrite** Alkaline phosphatase (ALP) Leukocytes Total bilirnbin (BILI) Clai·ity

Total protein Color Creatine Kinase Urobilinogen Bilirnbin NT-proBNP

For by-visit summai ies, visit windows as described in Section 4.2.2 will be used. In the case more than one result is collected for the same visit date the eai-liest result will be presented. For summaries across visits (e.g. maximum post-baseline value), scheduled, unscheduled and repeat assessments will be considered.

Abnornal laboratoly results ai e defined as any result outside the nonnal range (either below the lower limit of the nonnal range or above the upper limit of the nonnal range) at any visit

The following will be summai ized:

Reticulocyte Count

**MCV** 

MCH **MCHC** 

- A summaly of each laboratory pai ameter result and change from baseline by treatment group and visit
- A summaly of the number and percentage of subjects experiencing low, nonnal or high values at baseline and worst post-baseline result, by laboratoly paraineter and treatment group (shift table). Worst will be defined for both low and high abnonnalities for each pai ameter (i.e. each paraineter will be presented twice, once where low abno1malities ai·e worst and once where high abno1malities ai·e worst).
- A summary of the number and percentage of subjects experiencing at least one post-baseline laboratory abno1malities, by laboratory paraineter and treatment group. Both low and high abnonnalities will be repolied for each parameter.
- A summaiy of the number and percentage of subjects experiencing clinically significant laboratory abnolmalities, by laboratoly pai ameter, treatment group and visit and at any postbaseline visit

Clinically significant laboratory abnolmalities include laboratoly results of special interest and markers of potential liver injmy.

### Laboratory results of special interest:

- Hemoglobin < 8 g/dL or decrease > 2 g/dL from baseline
- Leukocytes  $< 4 \times 10^3/\mu L$
- Neutrophils  $< 1.0 \times 10^3/\mu L$
- Platelets  $< 30 \times 10^3/\mu L$

### Assessment of Liver Injury:

- ALT > 3x upper limit of normal (ULN)
- ALT > 5x ULN
- ALT > 10x ULN
- AST > 3x ULN
- AST > 5x ULN
- AST> 10x ULN
- ALP > 1.5x ULN
- BILI > 2x ULN
- ALT > 3x ULN and BILI > 2x ULN at the same visit
- AST > 3x ULN and BILI > 2x ULN at the same visit
- ALT or AST >3x ULN and BILI > 2x ULN at the same visit
- ALT > 3x ULN and BILI > 2x ULN and ALP < 2x ULN at the same visit
- AST > 3x ULN and BILI > 2x ULN and ALP < 2x ULN at the same visit
- ALT or AST >3x ULN and BILI > 2x ULN and ALP < 2x ULN at the same visit

By-subject listings of all laboratory data will be provided by treatment group, with abnormal values highlighted, and including center, subject identifier, age, sex, race, weight and visit. Laboratory reference ranges will also be listed.

Laboratory values (hematology, chemistry, coagulation/cardiac, and urinalysis) will be listed by subject and study time point including changes from baseline (with the exception of urinalysis).

All values outside the clinical reference ranges will be flagged in the data listings. The abnormal values will be flagged with 'L' for values below the lower limit of the clinical reference range and 'H' for values above the upper limit of the clinical reference range and included in the listings. Listings of abnormal or clinically significant results may be provided.

#### 4.9.4 Vital Signs, Physical Findings and Other Observations Related to Safety

The following vital sign parameters including change from baseline will be summarized by treatment group and visit for each study period.:

- Heart rate (HR: bpm)
- Respiratory rate (breaths per minute)
- Diastolic blood pressure (DBP; mmHg)
- Systolic blood pressure (SBP; mmHg)

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

• Body temperature (C)

fu addition, a summary of the number and percentage of patients meeting the following abno1mal vital sign criteria by visit and at any time during each study period:

- HR > 110 beats per minute
- HR > 20 beats per minute change from baseline
- DBP 90 mmHg
- DBP < 60 mmHg
- DBP > 20 mmHg change from baseline
- SBP 160 mmHg
- SBP < 90 mmHg
- SBP > 30 mmHg change from baseline

By-subject listings of vital sign parameters and physical examination results will be provided.

#### 4.9.5 Independent Data Monitoring Committee

An independent Data Monitoring Committee (DMC) will meet regularly while the study is ongoing and will be responsible for intel preting the results of both interim analyses.

Programs for analysis datasets and tables, listings, and figures (TLFs) for the DMC will be created by the blinded statistical team (biostatisticians and statistical programmers) using dummy randomization. These programs will be passed to the unblinded statistical team who will apply the true randomization. Blinded and unblinded directories will be maintained and access to the unblinded directory will be restricted to the unblinded team member until general study unblinding.

All TLFs (planned and ad hoc) created for the DMC will be developed following the guidelines defined in this SAP as appropriate.

Further details can be found in section 2 and in the DMC Charter.

**Table 4-3: Scheduled DMC Meetings** 

| Meetin!!: | Timin!!: | ReviewTvoe |
|---|---|---|
| 1 <sup>st</sup> Data Review<br>Meeting | After 10% of planned subjects are randomized, after 6 days of follow up post-first dose day, DMC will review the unblinded data for safety and change from baseline in clinically meaningful parameters such as change from baseline in hypoxemia measurements and the 7-point ordinal scale. | Safety |
| futerim Analysis 1<br>Meeting | After 22% of planned subjects have been treated and have completed 7 days of follow-up (i.e., completed the Day 15 Visit), the DMC will review unblinded accumulated data for safety and futility, including an analysis of whether any changes in measures of hypoxemia or oxygen saturation (e.g., SpOi/FiO2, PaO2/FiO2, | Safety/ Futility/ Change in oxygenation |

TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 Kinevant

KIN-1901-2001 Statistical Analysis Plan

| Meetine: | Timine: | Review Type |
|---|---|---|
| | or SpO2 on room air) are clinically meaningful. The DMC may recommend a pause in emolhnent at this time. | |
| futerim Analysis 2<br>Meeting | After 100 subjects completed the Day 29 Visit or died by Day 43 (Section 5.2.1), the DMC will review unblinded accumulated data. | Safety/ Superiority/Futility/<br>Sample Size Re-Estimation |
| 2 <sup>nd</sup> Data Review<br>Meeting (if<br>needed) | After 75% of planned subjects* are discharged from the hospital, complete the Day 43 Visit, discontinue the study early, or meet the primary mortality endpoint (by Day 43), the DMC will review unblinded accumulated data. | Safety |

#### 4.10 Other Analyses

#### 4.10.1 Pharmacokinetics

Sernm gimsilumab concentrations will be summarized (including geometric mean, CV%, and 95% confidence interval for post-baseline timepoints) at Baseline (pre-dose), Day 8 (pre-dose) and DoD/ET using descriptive statistics for the PK population. A scatter plot of individual concentrations (overlaid) versus actual time of sampling (relative to Day 1 dose) will be provided (conditioned on subjects receiving Day 1 or Day 1 and Day 8 dosesofstudy chug). Phannacokinetic data analysis will not be perfonned until after database lock as it is potentially unblinding.

Population PK analysis, if conducted, will be described in a separate analysis plan and report.

#### 4.10.2 Immunogenicity

Sernm anti-chug antibody (ADA) data will be summarized by visit and treatment for the safety analysis set (note, this analysis is distinct from the anti-GM-CSF auto-antibody test at Screening).

The following will be summai ized:

- ADA positive at baseline
- ADA negative post baseline
- ADA positive post baseline (regai dless of baseline; hnmunogenicity rate)
- ADA positive post baseline (but negative at baseline)

Assessment of ADA incidence and Day 8 pre-dose sernm gimsilumab concentration will be descriptively summarized by:

- ADA positive on any day
- ADA positive on Day 15

#### 4.10.3 Biomarker

Actual and change from baseline senun cytokines and safety biomarker SP-D results will be summarized by ti eatment at Baseline (pre-dose), Day 4, Day 8, and DoD/ET using descriptive statistics for the safety analysis set. Summary plots of actual and change from baseline sernm cytokines will be provided, where time=0 will be:

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant KIN-1901-2001 Statistical Analysis Plan

- Study Day 1
- Day of onset of symptoms

By-subject listings of biomarker results will be provided. Biomarker data analysis will not be performed until after database lock as it is potentially unblinding. Additional exploratory analyses may be performed.

### 4.11 Changes in the Conduct of the Study or Planned Analysis

SAP v3.0 incorporates changes to Interim Analysis 2 to include stopping criteria for superiority (Section 5.2.3) and to amend the stopping criteria for inferiority to use Mortality by Day 43 instead of Mortality by Day 29 (Section 5.2.4). SAP was updated before planned amendments to include these changes in the protocol and DMC Charter were finalized.

TP-GDO-WW-016-07.a **CONFIDENTIAL Project Document Version No. 4.0** Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019


Statistical Analysis Plan

#### 5 INTERIM ANALYSES

See also <u>Section 4.9.5</u> for infonnation on the DMC interim analyses. Please note the distinction between "DMC data review" and "DMC interim analysis".

#### 5.1 Interim Analysis 1

Objectives of interim analysis 1 (!Al) are for the DMC to

- review unblinded safety data
- · check efficacy for futility

### 5.1.1 Subjects to be included in interim analysis 1

Trigger date for !Al: 60 subjects ti-eated completed the Day 15 Visit or died

Subjects to be included in!Al: All subjects in the ITT analysis set randomized and treated at least 15 days prior to the!Al trigger date

#### 5.1.2 Analysis of efficacy endpoints at interim analysis 1

- Mortality up to Day 15: treatment effect estimated using CMH test strntified by baseline clinical status, odds ratio and 95% CI estimated using logistic regression model with treatment and baseline clinical status and independent variables.
- Overall survival: treatment effect estimated using logrank test, median, 25<sup>th</sup> percentile, 75<sup>th</sup> percentile smvival times in days, and by ti eatment surivival cmve as estimated using Kaplan-Meier methods.
- Alive and no mechanical ventilation on Day 15: ti-eatment effect estimated using CMH test sti-atified by baseline clinical status, odds ratio and 95% CI estimated using logistic regression model with ti-eatment and baseline clinical status and independent variables.
- Time to hospital discharge: ti-eatment effect estimated using logrank test, median, 25<sup>th</sup> percentile, 75<sup>th</sup> percentile smvival times in days, and by ti-eatment surivival cmve as estimated using Kaplan-Meier methods.
- Time to first 2-point improvement on 7-point ordinal scale: ti·eatment effect estimated using logrank test, median, 25<sup>th</sup> percentile, 75<sup>th</sup> percentile smvival times in days, and by ti·eatment surivival cmve as estimated using Kaplan-Meier methods.

#### 5.1.3 Futility criteria at interim analysis 1

No fonnal futility criteria were set. DMC met on June 19, 2020 and agreed that the study could continue without modification.

#### 5.2 Interim Analysis 2

Objectives of interim analysis 2 (IA2) are for the DMC to

- review unblinded safety data
- · check efficacy superiority stopping criteria
- check efficacy futility stopping criteria
- assess, if applicable, a sample size re-estimation based on the primary efficacy endpoint.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant

KIN-1901-2001 Statistical Analysis Plan

### 5.2.1 Subjects to be included in interim analysis 2

Trigger date for IA2: 100 subjects completed at least the Day 29 Visit (non-mortality data by Day 29) or died (moliality data by Day 43).

All subjects in the ITT analysis set randomized (and treated) at least 29 days prior to the IA2 trigger date and safety and efficacy data collected through the IA2 trigger date for these subjects will be included in the interim analysis.

Superiority analysis, futility analysis, and sample size re-estimation on the primary endpoint, Mo1iality by Day 43, will be based on subjects randomized (and treated) at least 43 days prior to the IA2 trigger date. Confinmation of survival status by Day 43 will consist of review of death date and eai·ly study withdrawal date by a clinical research associate and dates confinned by source data verification. If no death date is available site personnel should confinn whether or not the subject was still alive on Day 43.

### 5.2.2 Analysis of efficacy endpoints at interim analysis 2

The following efficacy endpoints will be analyzed at IA2:

- Mortality up to Day 43 as Estimand 1 described in Section 4.8.2
- Composite key secondary endpoint "Survival and no mechanical ventilation on Day 29" as described in Section 4.8.3.1.

#### 5.2.3 Superiority stopping criteria at interim analysis 2

The DMC may recommend stopping the study for superiority if the following condition is met:

D. Robust and compelling benefit of gimsilumab compaired to placebo on moliality up to Day 43, i.e., one-sided p-value < 0.0005.

### 5.2.4 Futility stopping criteria at interim analysis 2

The DMC may recommend stopping the study for futility, if at least one of the following conditions ai e met (relevant analysis specifications follow Section 5.2.1 and Section 5.2.2):

- No benefit of gimsilumab compared to placebo on m01iality up to Day 43, i.e., estimated treatment risk difference 0 and one-sided p-value 0.5.
- No benefit of gimsilumab compared to placebo on composite "survival and no mechnical ventilation on Day 29", i.e., estimated treatment response difference:::;0 and one-sided p-value 0.5.

### 5.2.5 Sample size re-estimation at interim analysis 2

If the study is neither stopped for superiority nor futility at IA2, the sample size will be re-assed by the following procedure for the primary efficacy endpoint moliality by Day 43:

- (A) The conditional power given the estimated common risk difference at IA2 will be calculated by
  - using the estimated common risk difference and its standai denor at IA2 (Estimand 1 described in Section 4.8.2)
  - assuming the cunent trend observed up to IA2 (stage 1) as hue disti·ibution pai·ameters for the remaining paii of the study (stage 2)
  - keeping the total sample size as 270 subjects.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Statistical Analysis Plan

- (B) If the conditional power is  $\geq 0.8$  (80%), then the initial sample size can be kept.
- (C) If the conditional power is < 0.8 (80%), then the sample size may be increased, so that
  - the conditional power calculated with the increased sample size is 0.8 (80%) for the final analysis combining the test statistics from first and second stage with pre-specified weights (<u>Cui/Hung/Wang 1999</u>) to maintain the type-I-error probability restricted to 0.025 one-sided; the two pre-specified weights are

$$w = \sqrt{\frac{n_1}{n_1}}$$
 with  $n$  denoting the number of subjects in the FAS for stage 1, i.e., subjects  $\frac{1}{27}$ 

randomized at least 43 days prior to the IA2 trigger date

$$w_2 = \sqrt{\frac{270 - n_1}{270}}$$
 where 270 –  $n_1$  represents the number of subjects in the FAS for stage 2,

i.e., subjects randomized 42 days prior to the IA2 trigger date or later

- but not increasing the maximum allowed total sample size of 400 subjects.
- (D) In order not disclosing too much information to sponsor and investigators, only the following categories for the total sample size can be recommended:
  - 270 subjects (i.e., no increase of the initial sample size)
  - 300 subjects
  - 330 subjects
  - 360 subjects
  - 400 subjects (i.e., the maximum allowed total sample size).

#### 5.2.6 Interim analysis 2 outcome

The DMC met on Aug 26<sup>th</sup>, 2020 to review results from interim analysis 2. After the meeting ad hoc analyses were requested to review efficacy endpoints by select subgroups and to perform some additional analyses on mechanical ventilation-free days. These analyses are documented in *KIN-1901-2001 PXL250621 Additional Statistical Analysis V1.0.docx*. Per sponsor decision, enrollment was stopped early with the intention of completing the study as planned for the 227 (84%) of subjects randomized on or before October 12, 2020. For planning purposes the ad hoc analyses were repeated using a data cut-off date of September 28, 2020 including all subjects randomized as of the cut-off date.

TP-GDO-WW-016-07.a CONFIDENTIAL
Effective Date: 30 Jan 19 Project Document
Related to: SOP-GDO-WW-019

Kinevant KIN-1901-2001

Statistical Analysis Plan

#### 6 REFERENCES

ARDS Definition Task Force. Ranieri VM, Rubenfield GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: The Berlin Definition. *JAMA*. 2012;307(23):2526-33

Beyersmann J, Allignol A, Schumacher M. Competing Risks and Multistate Models with R. Springer; 2012.

Cui L, Hung HMJ, Wang S-J. Modification of sample size in group sequential clinical trials. Biometric 1999;55:853-857

Ge M, et al. Covariate-adjusted difference in proportions from clinical trials using logistic regression and weighted risk differences. Drug Information Journal 2011;45:481-493

Liublinska V, Rubin DB. Sensitivity analysis for a partially missing binary outcome in a two-arm randomized clinical trial. Statistics in Medicine 2014;33:4170-4185

Yan X, Lee S, Li N. Missing data handling methods in medical device clinical trials. Journal of Biopharmaceutical Statistics 2009;19:1085-1098

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant KIN-1901-2001

Statistical Analysis Plan

**APPENDICES** 

**Project Document Version No.** 4.0 TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Effective Date: Date of last signature Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019


### 7.1 Schedule of Assessments

| | | | On-Treatment | |
|---|---|---|---|---|
| | Screen | Baseline <sup>a</sup> | Assessments<br>(only done if in hospital) | DoD / |
| Study Day (± Window) | -7 to 1 | 1 | Days 2 – 14, inclusive<br>(All ± 1 day) | - |
| Week | 0 | 0 | 1 to 2 | 0-6 |
| Informed consent and randomization | X | | | |
| Inclusion/Exclusion criteria | X | Хр | | |
| Demographic information, medical history, prior medications° | X | | | |
| Local QuantiFERON® test⁴ | X | | | |
| Local Viral Screen (HBsAG, HCV RNA/Ag, HIV)d | X | | | |
| Height and Weighte | X | | | |
| Local Urine pregnancy test β-hCG and follicle-stimulating hormone (women only) <sup>f</sup> | X | | | |
| Central sample for anti-GM-CSF autoAba (result not required for determination of eligibility) | X | | | |
| Chest X-ray or chest CT scan (within 3 days of Day 1) | X | | | |
| Local qualitative sample (e.g., nasopharyngeal swab) for PCR SARS-CoV-2 (if not already documented) | X | | | |
| Central quantitative sample (e.g., nasopharyngeal swab) for PCR SARS-CoV-29 | | X | Days 2 and 9 | X |
| Physical examination <sup>h</sup> and vital signs (blood pressure, heart rate, respiration rate, and body temperature) <sup>i</sup> | X | X | Daily, only while hospitalized | X |
| Central clinical laboratory measurements (hematology, blood chemistry [including CRP, ferritin, LDH, procalcitonin, troponin I], coagulation [including D-dimer], and urinalysis) <sup>i</sup> | X | х | Days 4 and 8 | X |
| Administration of IV study drug <sup>k</sup> | 0 | X | Day 8 | |
| Central PK samples for quantification of gimsilumab serum concentration | | Predose | Predose on Day 8 | X |
| Central samples for cytokine panel | 0 | X | Days 4 and 8 | X |

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0
Effective Date: 30 Jan 19
Related to: SOP-GDO-WW-019


| Schedule of Assessments: Screening and Treatment Period | | | | |
|---|---|---|---|---|
| | Screen | Baselinea | On-Treatment<br>Assessments<br>(only done if in hospital) | DoD / |
| Study Day (± Window) | -7 to 1 | 1 | Days 2 – 14, inclusive<br>(All ± 1 day) | - |
| Week | 0 | 0 | 1 to 2 | 10-01 |
| Central samples for SP-D measurement | | X | Day 8 | X |
| Central sample for immunogenicity (antibodies to gimsilumab) | | X | | X |
| 7-point Ordinal Scale | | X | Daily, only while hospitalized | Х |
| National Early Warning Score (NEWS) | | X | Daily, only while hospitalized | X |
| SOFA score | | X | Daily, only while in ICU | X |
| SpO <sub>2</sub> /FiO <sub>2</sub> , and if performed, PaO <sub>2</sub> /FiO <sub>2</sub> (can be imputed) | Х | X | Daily, only while hospitalized | X |
| Oxygenation requirements | X | X | Daily, only while hospitalized | Х |
| Ventilation requirements <sup>1</sup> | Х | X | Daily, only while hospitalized | X |
| ECMO requirements | | X | Daily, only while hospitalized | Х |
| Concomitant medications/concurrent procedures <sup>m</sup> | | X | Daily, only while hospitalized | X |
| Adverse event monitoring <sup>n</sup> | | X | Daily, only while hospitalized | X |

β-hCG = beta human chorionic gonadotropin; anti-GM-CSF autoAb = anti-granulocyte macrophage colony- stimulating factor auto-antibody; DoD = Day of Discharge from hospital; ECMO = extracorporeal membrane oxygenation; EoS = End-of-Study; ET = early termination; FiO<sub>2</sub> = fraction of inspired oxygen; HBsAg = hepatitis B surface antigen; HCVAb = hepatitis C virus antibodies; HIV = human immunodeficiency virus; ICU = Intensive Care Unit; IGRA = interferon gamma release assay; IV = intravenous; PCR = polymerase chain reaction; PK = pharmacokinetics; SOFA = sequential organ failure assessment; SP-D = serum surfactant protein D; SpO<sub>2</sub> = peripheral capillary oxygen saturation

- a. Baseline assessments should be performed prior to study drug administration. Assessments performed within 48 hours of Baseline do not need to be repeated at Baseline.
- b. Verification that no changes affecting eligibility have occurred since Screening will be performed at the Baseline/Day 1 Visit.
- c. Collect medication history from the 30 days leading up to, and including, the time of the Screening Visit, including date of onset of COVID-19 symptoms, prescription medications, over-the-counter medications, and herbal supplements/vitamins.
- d. Sample will be collected, but enrollment can continue without receiving results first. HCV testing can be RNA or Ag, only to confirm suspected infection. If a subject is diagnosed with latent TB (positive QuantiFERON Gold or purified protein derivative [PPD]), hepatitis B or C, or HIV during the study, the Investigator must discuss this with the medical monitor and a decision will then be made concerning the second dose of gimsilumab, if applicable. In the event the QuantiFERONn Gold assay is not available, and the site performs a different IGRA such as T Spot, then the alternative IGRA will be acceptable for patient screening and enrollment. Enrollment should not be delayed to obtain the QuantiFERONn Gold assay in lieu of the IGRA available at the site. If no IGRA test is available, PPD can be used.
- e. Height will be assessed only once (at Screening). Estimated height and weight are acceptable if unable to be measured due to patient clinical condition.
- f. The Screening sample can be assessed using local laboratory services for Screening/Eligibility purposes.

TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


#### Kinevant

KIN-1901-2001 Statistical Analysis Plan

- q. When at all possible, if only 1 nostril is swabbed for viral assessments, the same nostril should be used for all subsequent samples.
- An abbreviated, targeted physical examination will be performed based on the subject's clinical status and what the clinic staff feel is appropriate.
- Vital signs will be assessed at all timepoints specified above. On study drug administration days, vital signs will be assessed pre-dose (within 15 minutes) and ± 30 minutes post end of
- j. ALT, AST, CRP, and Ferritin can be assessed using local laboratory services for Screening. For all on-study laboratory assessments, if central laboratory assessments cannot be collected for any reason, best efforts will be made to record local laboratory data.
- k. Subjects will receive a single IV infusion of blinded study treatment on Day 1 and Day 8. The Day 8 dose will be omitted if the subject is discharged or is no longer in need of supplemental oxygen or ventilatory support for >48 hours.
- If subject is receiving mechanical ventilation, the following parameters will be recorded: type of ventilation (CPAP, BiPAP, or intubation), FiO2, SpO2, ventilation rate, pulse, tidal volume, positive end-expiratory pressure (PEEP), and airway pressure.
- m. Collect information on concomitant medications and concurrent procedures from the time of informed consent through the EoS Visit (or ET Visit if subject discontinues early), including prescription medications, over-the-counter medications, and herbal supplements/vitamins.
- Adverse event monitoring will include assessment of treatment-emergent AEs (TEAEs), serious adverse events (SAEs), and severe AEs (Grade 3 or 4 events).

Note: SCREENING LABORATORY ASSESSMENTS: For all screening laboratory assessments, if more than one result is available during the screening period, the most recent value will be used as the screening value and for determination of eligibility.

Note: All subjects who are discharged from the hospital will undergo all Day-of-Discharge (DoD) Visit assessments; daily in-hospital assessments will only need to be performed once on DoD. All subjects who discontinue from the study prematurely will undergo all Early Termination (ET) Visit assessments, whenever possible. All subjects who discontinue treatment and/or the study early will be followed for Day 43 all-cause mortality.

TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No. 4.0** Effective Date: 30 Jan 19 **Project Document Effective Date:** Date of last signature Related to: SOP-GDO-WW-019 

| Schedul<br>(Visits will be in-hosp | | | ollow-up Pe<br>ubject has l | | rged) | | | |
|---|---|---|---|---|---|---|---|---|
| Study Day (± Window) | 15<br>(± 2) | 22<br>(± 2) | 29<br>(± 2) | 36<br>(± 2) | 43°<br>(± 2) | 85<br>(± 2) | EoS<br>169<br>(± 2) | DoD / |
| Week | 2 | 3 | 4 | 5 | 6 | 12 | 24 | , s <del></del> |
| Procedures/Assessments | 10 | | | | | | | • |
| SOFA Score | | Daily, onl | y if in ICU, t | hrough Day 4 | 13 | 8 8<br>6 8 | | X |
| National Early Warning Score (NEWS) | Da | ily, only wh | ile hospitaliz | zed, through [ | Day 43 | | | X |
| Central samples for cytokine panel Hosp Hosp | | | | | | 58 | | |
| Central samples for SP-D measurement | | | Hosp | | | | | |
| Central sample for immunogenicity (antibodies to gimsilumab) | Hosp | | Hosp | | Hosp | | | |
| Central clinical laboratory measurements (hematology, blood chemistry [including CRP, ferritin, LDH, procalcitonin, troponin I], coagulation [including D-dimer], and urinalysis) <sup>b</sup> | | Hosp | Hosp | Hosp | Hosp | | | х |
| SpO <sub>2</sub> /FiO <sub>2</sub> , and if performed, PaO <sub>2</sub> /FiO <sub>2</sub> (can be imputed) | Da | ily, only wh | ile hospitaliz | zed, through [ | Day 43 | | | X |
| Oxygenation requirements | Dai | ly, only whi | le hospitaliz | ed, through [ | ay 43: | | | X |
| Ventilation requirements | Da | ily, only wh | ile hospitaliz | zed, through [ | Day 43 | | | X |
| ECMO requirements | Daily, only while hospitalized, through Day 43 | | | | X | | | |
| Concomitant medications/concurrent procedures | Daily, only while hospitalized | | | X | X | X | | |
| Physical examination and vital signs (blood pressure, heart rate, respiration rate, and body temperature) | | Hosp | Hosp | Hosp | Hosp | | | Х |
| 7-point Ordinal Scale Daily, only while hospitalized, through Da | | | ay 43ª | X | Х | X | | |
| Adverse event monitoring <sup>e</sup> | Daily, only while hospitalized | | | | X | X | X | |

ECMO = extracorporeal membrane oxygenation; EoS = End-of-Study; FiO<sub>2</sub> = fraction of inspired oxygen; Hosp = Assessment to be performed only if subject has not been discharged; ICU = Intensive Care Unit; SOFA = sequential organ failure assessment; SP-D = serum surfactant protein D; SpO<sub>2</sub> = peripheral capillary oxygen saturation

- a. Day 43 will be used for the primary all-cause mortality endpoint.
- b. For all on-study laboratory assessments, if central laboratory assessments cannot be collected for any reason, best efforts will be made to record local laboratory data.
- c. IF DISCHARGED, will be measured via phone follow-up on Day 15, 22, 29, 36, and 43.
- d. IF DISCHARGED, will be measured via phone follow-up on Day 15, 22, 29, 36, 43, 85, and 169.
- e. Adverse event monitoring will include assessment of treatment-emergent AEs (TEAEs), serious adverse events (SAEs), and severe AEs (Grade 3 or 4 events)

Note: Assessments at time points indicated with "Hosp" will only be conducted if the subject has not yet been discharged from the hospital. Assessments indicated with an 'X' will be performed in-hospital if the subject has not been discharged or via phone if subject has been discharged from the hospital.

Note: All subjects who are discharged from the hospital will undergo all Day-of-Discharge (DoD) Visit assessments; daily in-hospital assessments will only need to be performed once on DoD. All subjects who discontinue from the study prematurely will undergo all Early Termination (ET) Visit assessments, whenever possible.

All subjects who discontinue treatment and/or the study early will be followed for Day 43 all-cause mortality.

TP-GDO-WW-016-07.a Effective Date: 30 Jan 19

**CONFIDENTIAL** 

Project Document Version No. 4.0

**Project Document Effective Date**: Date of last signature


Related to: SOP-GDO-WW-019

## 7.2 Adverse Events of Special Interest


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant


TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


K.inevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL

**Project Document Version No.** 4.0 Project Document Effective Date: Date of last signature


Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant KIN-1901-2001

Statistical Analysis Plan


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant KIN-1901-2001

Statistical Analysis Plan


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0

Project Document Effective Date: Date of last signature


Statistical Analysis Plan

Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Statistical Analysis Plan

Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Statistical Analysis Plan

Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature

Kinevant KIN\_1901\_2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

IAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a CONFIDENTIAL Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019

**Project Document Version No.** 4.0


Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant KIN-1901-2001

Statistical Analysis Plan


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant KIN\_1901\_2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

IAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


K.inevant KIN-1901-2001

| Statistical | Analy | vsis | Plan |
|-------------|-------|-------|-------|
| Statistical | Amar | y 515 | 1 1ai |


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL

**Project Document Version No.** 4.0

**Project Document Effective Date:** Date of last signature


K.inevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


K.inevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


K inevant

NaITow

NaITow

NaITow

Broad

Broad

Broad

A

A

A

A

A

A


TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No. 4.0** Project Document Effective Date: Date of last signature Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 

Platelet production decreased

Megakarvocvtes abnonnal

Platelet count abno1mal

Platelet toxicity

Platelet disorder

Thrombocytopenia

10035540

10059440

10043554

10027118

10035526

10035532

K.inevant KIN-1901-2001

| Statistical | Analy | 7010 | Plan |
|-------------|-------|------|------|
| Statistical | Allar | VSIS | ГІап |


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant KIN\_1901\_2001


TP-GDO-WW-016-07.a CONFIDENTIAL Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

 $\textbf{Project Document Version No.}\ 4.0$ **Project Document Effective Date**: Date of last signature


Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant


TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 4.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature 

Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant KIN-1901-2001

Statistical Analysis Plan


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


K.inevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL

Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 4.0
Project Document Effective Date: Date of last signature


Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

**Project Document Version No.** 4.0 CONFIDENTIAL **Project Document Effective Date**: Date of last signature

Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 122

**Project Document Version No.** 4.0 CONFIDENTIAL **Project Document Effective Date**: Date of last signature

Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

**Project Document Version No.** 4.0 CONFIDENTIAL **Project Document Effective Date**: Date of last signature

Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

**Project Document Version No.** 4.0 CONFIDENTIAL Project Document Effective Date: Date of last signature

Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

**Project Document Version No.** 4.0 CONFIDENTIAL **Project Document Effective Date**: Date of last signature

Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

**Project Document Version No.** 4.0 CONFIDENTIAL **Project Document Effective Date**: Date of last signature

Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

**Project Document Version No.** 4.0 CONFIDENTIAL **Project Document Effective Date**: Date of last signature

Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

**Project Document Version No.** 4.0 CONFIDENTIAL **Project Document Effective Date**: Date of last signature
Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

**Project Document Version No.** 4.0 CONFIDENTIAL **Project Document Effective Date**: Date of last signature

K.inevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL **Project Document Version No. 4.0** 

Project Document Effective Date: Date oflast signature Page 109 of

Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

**Project Document Version No.** 4.0 CONFIDENTIAL **Project Document Effective Date**: Date of last signature

Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

**Project Document Version No.** 4.0 CONFIDENTIAL Project Document Effective Date: Date of last signature

Hypotension

Biliary fibrosis

Hypotensive crisis

Post procedural hypotension

K.inevant KIN-1901-2001

Broad

Broad Broad D

D

D


Statistical Analysis Plan

10021097

10083659

10084013


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

A


Project Document Effective Date offset signature

**Project Document Effective Date:** Date oflast signature


10004664

Nanow

Kinevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 122

**Project Document Version No.** 4.0 CONFIDENTIAL Project Document Effective Date: Date of last signature


Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

Project Document Effective Date: Date of last signature

ed to: SOP-GDO-WW-019 Page 114 of

K.inevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

**Project Document Version No.** 4.0 CONFIDENTIAL Project Document Effective Date: Date of last signature

K.inevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

Project Document Effective Date: Date of last signature

K.inevant KIN-1901-2001

Statistical Analysis Plan


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

**Project Document Version No.** 4.0 CONFIDENTIAL Project Document Effective Date: Date of last signature

Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

**CONFIDENTIAL Project Document Version No.** 4.0 **Project Document Effective Date**: Date of last signature


K.inevant KIN-1901-2001


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

**Project Document Version No.** 4.0 CONFIDENTIAL Project Document Effective Date: Date of last signature

Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

Project Document Effective Date: Date of last signature

o: SOP-GDO-WW-019 Page 120 of


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 **CONFIDENTIAL Project Document Version No.** 4.0 **Project Document Effective Date**: Date of last signature


Kinevant


TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

122

Project Document Effective Date: Date of last signature


## Signature Page for VV-TMF-311484 vl.0

| Reason for signing: Approved | Name: Role: Date re: 14-Nov-2020 23:32:38 GMT+0000 |
|---|---|
| Reason for signing: Approved | 16-Nov-2020 14:45:55 GMT+0000 |
| Reason for signing: Approved | re: 17-Nov-2020 01:30:32 GMT+0000 |
| Reason for signing: Approved | 17-Nov-2020 12:43:53 GMT+0000 |

Signature Page for VV-TMF-311484 vl.0